CLINICAL TRIAL: NCT01272037
Title: A Phase III, Randomized Clinical Trial of Standard Adjuvant Endocrine Therapy +/- Chemotherapy in Patients With 1-3 Positive Nodes, Hormone Receptor-Positive and HER2-Negative Breast Cancer With Recurrence Score (RS) of 25 or Less. RxPONDER: A Clinical Trial Rx for Positive Node, Endocrine Responsive Breast Cancer
Brief Title: Tamoxifen Citrate, Letrozole, Anastrozole, or Exemestane With or Without Chemotherapy in Treating Patients With Invasive RxPONDER Breast Cancer
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2011-02623; NCI-2011-02623 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); S12-03603; CDR0000692475; PS1007_A11PAMDREVW01; SWOG-S1007; S1007 (Other: SWOG); S1007 (Other: CTEP); U10CA032102 (NIH); U10CA180830 (NIH); U10CA180888 (NIH)
Record Dates: First submitted 2011-01-06; First posted 2011-01-07 (Estimated); Results first posted 2023-06-27 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-10

CONDITIONS: Breast Ductal Carcinoma In Situ; Invasive Breast Carcinoma; Multicentric Breast Carcinoma; Multifocal Breast Carcinoma; Synchronous Bilateral Breast Carcinoma
MeSH Terms: conditions — Carcinoma, Intraductal, Noninfiltrating | interventions — Anastrozole; exemestane; Letrozole; Neoadjuvant Therapy; Tamoxifen

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm I (chemotherapy and endocrine therapy) (Experimental): Patients receive a protocol-approved chemotherapy regimen based on the patient and/or physician preference. Patients then receive a protocol-approved adjuvant endocrine therapy comprising tamoxifen citrate, an aromatase inhibitor (anastrozole, letrozole, or exemestane), or both for 5-10 years in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Anastrozole; Drug: Exemestane; Other: Laboratory Biomarker Analysis; Drug: Letrozole; Other: Quality-of-Life Assessment; Drug: Systemic Chemotherapy; Drug: Tamoxifen Citrate
- Arm II (endocrine therapy) (Experimental): Patients receive a protocol-approved endocrine therapy comprising tamoxifen citrate, an aromatase inhibitor (anastrozole, letrozole, or exemestane), or both for 5-10 years in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Anastrozole; Drug: Exemestane; Other: Laboratory Biomarker Analysis; Drug: Letrozole; Other: Quality-of-Life Assessment; Drug: Tamoxifen Citrate

INTERVENTIONS:
Drug: Anastrozole — Given PO
  Other Names: Anastrazole; Arimidex; ICI D1033; ICI-D1033; ZD-1033
Drug: Exemestane — Given PO
  Other Names: Aromasin; FCE-24304
Other: Laboratory Biomarker Analysis — Correlative studies
Drug: Letrozole — Given PO
  Other Names: CGS 20267; CGS-20267; CGS20267; Femara; Fempro
Other: Quality-of-Life Assessment — Ancillary studies (closed as of 12/1/12)
  Other Names: Quality of Life Assessment
Drug: Systemic Chemotherapy — Given IV
  Arms: Arm I (chemotherapy and endocrine therapy)
Drug: Tamoxifen Citrate — Given PO
  Other Names: Apo-Tamox; Clonoxifen; Dignotamoxi; Ebefen; Emblon; Estroxyn; Fentamox; Gen-Tamoxifen; Genox; ICI 46,474; ICI 46474; ICI-46474; ICI46474; Jenoxifen; Kessar; Ledertam; Lesporene; Nolgen; Noltam; Nolvadex; Nolvadex-D; Nourytam; Novo-Tamoxifen; Novofen; Noxitem; Oestrifen; Oncotam; PMS-Tamoxifen; Soltamox; TAM; Tamax; Tamaxin; Tamifen; Tamizam; Tamofen; Tamoxasta; Tamoxifeni Citras; Zemide

SUMMARY:
This randomized phase III clinical trial studies how well tamoxifen citrate, anastrozole, letrozole, or exemestane with or without chemotherapy work in treating patients with breast cancer that has spread from where it began in the breast to surrounding normal tissue (invasive). Estrogen can cause the growth of breast cancer cells. Hormone therapy, using tamoxifen citrate, may fight breast cancer by blocking the use of estrogen by the tumor cells. Aromatase inhibitors, such as anastrozole, letrozole, and exemestane, may fight breast cancer by lowering the amount of estrogen the body makes. Drugs used in chemotherapy work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. It is not yet known whether giving tamoxifen citrate, anastrozole, letrozole, or exemestane is more effective with combination chemotherapy in treating patients with breast cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To determine the effect of chemotherapy in patients with node positive breast cancer who do not have high recurrence scores (RS) by Oncotype DX.

SECONDARY OBJECTIVES:

I. To compare overall survival (OS), distant disease-free survival (DDFS) and local disease-free interval (LDFI) by receipt of chemotherapy or not and its interaction with RS.

II. To compare the toxicity across the treatment arms. III. To perform other molecular assays or test other signatures that measure prognosis and potential benefit of chemotherapy and compare them to Oncotype DX.

IV. To determine the impact of management with Oncotype DX on patient-reported anxiety (co-primary Health-Related Quality of Life [HRQL] outcome) prior to screening, after disclosure of test results, and during the randomized trial.

V. To determine the impact of Oncotype DX on the initial management cost of node-positive, hormone receptor (HR)-positive, human epidermal growth factor receptor 2 (HER2)-negative breast cancer.

VI. To compare patient-reported utilities (e.g., quality of life [QOL]) for those randomized to chemotherapy versus no chemotherapy.

VII. Using modeling and DFS information from the trial, to estimate the cost-effectiveness of management with Oncotype DX vs usual care.

VIII. To determine the role of other assays as predictors of DFS, DDFS, and LDFI for patients randomized to chemotherapy versus no chemotherapy.

IX. To determine the impact of treatment with chemotherapy versus no chemotherapy on patient-reported fatigue and cognitive concerns (secondary HRQL outcomes).

X. To determine the impact of management with Oncotype DX on patient-reported decision conflict, perceptions regarding Oncotype DX testing, and survivor concerns prior to screening, after disclosure of test results, and during the randomized trial (secondary HRQL outcomes).

XI. The presence of circulating tumor cells (CTC+) using two CTC platforms will be assessed at up to two time points to assess late recurrence in those still at risk for the primary outcome.

XII. To compare clinically reported menopausal status with status categorized by serum hormone levels determined from baseline serum in women under age 55 years and to assess subsequent association with outcomes.

BANKING OBJECTIVE:

I. To bank specimens for future correlative studies.

OUTLINE: Patients are randomized to 1 of 2 treatment arms.

ARM I: Patients receive a protocol-approved chemotherapy regimen based on the patient and/or physician preference. Patients then receive a protocol-approved adjuvant endocrine therapy comprising tamoxifen citrate, an aromatase inhibitor (anastrozole, letrozole, or exemestane), or both for 5-10 years in the absence of disease progression or unacceptable toxicity.

ARM II: Patients receive a protocol-approved endocrine therapy comprising tamoxifen citrate, an aromatase inhibitor (anastrozole, letrozole, or exemestane), or both for 5-10 years in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 3 months for 1 year, every 6 months for 4 years, and then yearly for 15 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have a histologically confirmed diagnosis of node positive (1-3 nodes) invasive breast carcinoma with positive estrogen and/or progesterone receptor status, and negative HER-2 status; estrogen and progesterone receptor positivity must be assessed according to American Society of Clinical Oncology (ASCO)/College of American Pathologists (CAP) guidelines as either estrogen receptor (ER) or progesterone receptor (PR) >= 1% positive nuclear staining; HER-2 test result negativity must be assessed as per ASCO/CAP 2013 guidelines using immunohistochemistry (IHC), in situ hybridization (ISH) or both; HER-2 is negative if a single test (or all tests) performed in a tumor specimen show: a) IHC negative (0 or 1+) or b) ISH negative using single probe or dual probe (average HER-2 copy number < 4.0 signals per cell by single probe or HER-2/CEP ration < 2.0 with an average copy number < 4.0 signals per cell by dual probe); if HER-2 IHC is 2+, evaluation for gene amplification (ISH) must be performed and the ISH must be negative; ISH is not required if IHC is 0 or 1+; HER-2 equivocal is not eligible
* Patients with multifocal, multicentric and synchronous bilateral breast cancers are allowed

  * Multifocal disease is defined as more than one invasive cancer < 2 cm from the largest lesion within the same breast quadrant; (NOTE: the Oncotype DX testing must be completed on the largest lesion)
  * Multicentric disease is defined as more than one invasive cancer >= 2 cm from the largest lesion within the same breast quadrant or more than one lesion in different quadrants (NOTE: Oncotype DX testing should be completed on all tumors and the determination for eligibility should be made on the highest recurrence score)
  * Synchronous bilateral disease is defined as invasive breast cancer with positive lymph nodes (axillary or intramammary) in at least one breast, diagnosed within 30 days of each other; (NOTE: the Oncotype DX testing should be completed on both tumors and the tumor with the highest recurrence score should be used)
* Patients will have undergone axillary staging by sentinel node biopsy or axillary lymph nodes dissection (ALND); patients must have at least one, but no more than three known positive lymph nodes (pN1a, pN1b or pN1c); patients with micrometastases as the only nodal involvement (pN1mi) are not eligible; patients with positive sentinel node are not required to undergo full axillary lymph node dissection; this is at the discretion of the treating physician; axillary node evaluation is to be performed per the standard of care at each institution
* Patients with a prior diagnosis of contralateral ductal carcinoma in situ (DCIS) are eligible if they underwent a mastectomy or lumpectomy with whole breast radiation; prior partial breast irradiation, including brachytherapy, is not allowed; patients with a prior diagnosis of ipsilateral DCIS or invasive breast cancer who received radiation to that breast are not eligible
* Patients must have had either breast-conserving surgery with planned radiation therapy or total mastectomy (with or without planned postmastectomy radiation); patients must have clear margins from both invasive breast cancer and DCIS (as per local institutional guidelines); lobular carcinoma in situ (LCIS) at the margins is allowed
* Registration of patients who have not yet undergone Oncotype DX screening must occur no later than 56 days after definitive surgery; (for all patients, Step 2 Registration must occur within 84 days after definitive surgery); if the Oncotype DX Breast Cancer Assay has not been performed, patients must be willing to submit tissue samples for testing to determine the Recurrence Score value; a representative block or unstained sections from the representative block are sent directly to Genomic Health for Oncotype DX Breast Cancer Assay which will be performed according to the standard commercial process

  * If the Oncotype DX Recurrence Score is already known and is 25 or less, the patient must be registered to Step 2 immediately following Step 1 registration; if the Oncotype DX Recurrence Score is already known and is greater than 25, the patient is ineligible
* Patients must be females >= 18 years of age. As the Oncotype DX recurrence score has not been validated in men with breast cancer, men are not eligible for this study
* Patients must have a complete history and physical examination within 28 days prior to registration
* Patients must have a performance status of 0-2 by Zubrod criteria
* Patients must be able to receive taxane and/or anthracycline based chemotherapy
* Patients must not have received an aromatase inhibitor (AI) or a selective estrogen receptor modulator (SERM) such as tamoxifen or raloxifene within 5 years prior to registration
* No other prior malignancy is allowed except for adequately treated basal cell (or squamous cell) skin cancer, in situ cervical cancer, or other cancer for which the patient has been disease-free for 5 years
* The Quality of Life and Economic Substudy is permanently closed to accrual effective 12/1/12; patients who consented to QOL prior to 12/1/12 should continue to complete QOL forms per their expectation report; patients who are able to complete a questionnaire in English must be offered the opportunity to participate in the Quality of Life and Economic Substudy; (The Quality of Life and Economic Substudy is available to U.S. INSTITUTIONS ONLY); patients who are not able to complete a questionnaire in English are registered to S1007 without participating in the Quality of Life and Economic Substudy

  * Patients who consent to participate in the Quality of Life and Economic Substudy and who do not yet know the results of their Oncotype DX screening must agree to complete the S1007 Health-Related Quality of Life Questionnaire: Enrollment between 14 days prior to and 7 days after Step 1 Registration
  * Patients who consent to participate in the Quality of Life and Economic Substudy and who do already know their Oncotype DX Recurrence Score (and it is 25 or less) will proceed to Step 2 Registration without completing the S1007 Health-Related Quality of Life Questionnaire Enrollment Form (but will complete the S1007 Health-Related Quality of Life Questionnaire: Randomized Study Form)
* Patients or their legally authorized representative must be informed of the investigational nature of this study and must sign and give written informed consent in accordance with institutional and federal guidelines; for Step 1 registration of patients who have not yet submitted specimens for the Oncotype DX Breast Cancer Assay, the appropriate consent form is the Step 1 Consent Form; for both Step 1 and Step 2 registration of patients whose Recurrence Score is already known and is 25 or less, the appropriate consent form is the Step 2 Consent Form
* As a part of the Oncology Patient Enrollment Network (OPEN) registration process the treating institution's identity is provided in order to ensure that the current (within 365 days) date of institutional review board approval for this study has been entered in the system
* STEP 2 REGISTRATION
* Recurrence score (RS) by Oncotype DX must be =< 25
* Step 2 Registration must take place within 84 days after definitive surgery; patients must not have begun chemotherapy or endocrine therapy for their breast cancer prior to randomization
* Patients randomized to either arm may also co-enroll in phase III trials that compare local therapies, or compare systemic therapies (such as chemotherapy, if randomized to Arm I of S1007)
* The Quality of Life and Economic Substudy is permanently closed to accrual effective 12/1/12; patients at U.S. INSTITUTIONS who consent to participate in the Quality of Life and Economic Substudy must agree to complete the S1007 Health-Related Quality of Life Questionnaire: Randomized Study Form after Recurrence Score results and randomized treatment status are known but before treatment has been initiated
* Patients or their legally authorized representative must be informed of the investigational nature of this study and must sign and give written informed consent in accordance with institutional and federal guidelines; for all patients the appropriate consent form for this registration is the Step 2 Consent
* STEP 3 REGISTRATION CBALR TM Substudy
* Patients must be disease-free, with no prior invasive recurrence at time of registration to Step 3
* Patients must be registered to Step 3 no more than 8 years after randomization (Step 2 Registration) and must agree to have samples drawn within 28 days after registration to Step 3
* Patients must agree to have blood samples collected at up to 3 timepoints: 1) within 28 days after registration to Step 3, 2) 2-3 years after time of registration to Step 3, and 3) At time of invasive recurrence (if applicable). Patients must also agree to have tissue submitted at time of invasive recurrence (if applicable) from the invasive recurrence biopsy (where tissue is available)

Exclusion Criteria:

* Patients must not have inflammatory breast cancer and must not have metastatic disease
* Patients must not have begun chemotherapy or endocrine therapy for their breast cancer prior to registration
* Patients must not require chronic treatment with systemic steroids (inhaled steroids are allowed) or other immunosuppressive agents
* Patients must not be pregnant or nursing; women of reproductive potential must have agreed to use an effective contraceptive method; a woman is considered to be of "reproductive potential" if she has had menses at any time in the preceding 12 consecutive months; in addition to routine contraceptive methods, "effective contraception" also includes heterosexual celibacy and surgery intended to prevent pregnancy (or with a side-effect of pregnancy prevention) defined as a hysterectomy, bilateral oophorectomy or bilateral tubal ligation; however, if at any point a previously celibate patient chooses to become heterosexually active during the time period for use of contraceptive measures outlined in the protocol, he/she is responsible for beginning contraceptive measures

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5018 (Actual)
Dates: Start 2011-01-15 (Actual); Primary Completion 2023-02-01 (Actual); Study Completion 2032-10-01 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Kevin M Kalinsky, Principal Investigator — SWOG Cancer Research Network
Locations (1572):
- United States (1439):
  - Northeast Alabama Regional Medical Center, Anniston, Alabama
  - University of Alabama at Birmingham Cancer Center, Birmingham, Alabama
  - Providence Hospital, Mobile, Alabama
  - University of South Alabama Mitchell Cancer Institute, Mobile, Alabama
  - Anchorage Associates in Radiation Medicine, Anchorage, Alaska
  - Anchorage Radiation Therapy Center, Anchorage, Alaska
  - Alaska Breast Care and Surgery LLC, Anchorage, Alaska
  - Alaska Oncology and Hematology LLC, Anchorage, Alaska
  - Alaska Regional Hospital, Anchorage, Alaska
  - Alaska Women's Cancer Care, Anchorage, Alaska
  - Anchorage Oncology Centre, Anchorage, Alaska
  - Katmai Oncology Group, Anchorage, Alaska
  - Providence Alaska Medical Center, Anchorage, Alaska
  - Fairbanks Memorial Hospital, Fairbanks, Alaska
  - Virginia G Piper Cancer Care-Del Camino, Scottsdale, Arizona
  - Mercy Hospital Fort Smith, Fort Smith, Arkansas
  - CHI Saint Vincent Cancer Center Hot Springs, Hot Springs, Arkansas
  - NEA Baptist Memorial Hospital and Fowler Family Cancer Center - Jonesboro, Jonesboro, Arkansas
  - NEA Baptist Memorial Hospital, Jonesboro, Arkansas
  - Kaiser Permanente-Anaheim, Anaheim, California
  - East Bay Medical Oncology Hematology Medical Associates-Antioch, Antioch, California
  - Kaiser Permanente-Deer Valley Medical Center, Antioch, California
  - PCR Oncology, Arroyo Grande, California
  - Sutter Auburn Faith Hospital, Auburn, California
  - Sutter Cancer Centers Radiation Oncology Services-Auburn, Auburn, California
  - Kaiser Permanente-Baldwin Park, Baldwin Park, California
  - Kaiser Permanente-Bellflower, Bellflower, California
  - Alta Bates Summit Medical Center-Herrick Campus, Berkeley, California
  - Providence Saint Joseph Medical Center/Disney Family Cancer Center, Burbank, California
  - Mills-Peninsula Medical Center, Burlingame, California
  - Sutter Cancer Centers Radiation Oncology Services-Cameron Park, Cameron Park, California
  - Mercy San Juan Medical Center, Carmichael, California
  - East Bay Radiation Oncology Center, Castro Valley, California
  - Eden Hospital Medical Center, Castro Valley, California
  - Valley Medical Oncology Consultants-Castro Valley, Castro Valley, California
  - Community Cancer Institute, Clovis, California
  - University Oncology Associates, Clovis, California
  - John Muir Medical Center-Concord, Concord, California
  - UC Irvine Health Cancer Center-Newport, Costa Mesa, California
  - Sutter Davis Hospital, Davis, California
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - Epic Care-Dublin, Dublin, California
  - Bay Area Breast Surgeons Inc, Emeryville, California
  - Epic Care Partners in Cancer Care, Emeryville, California
  - Kaiser Permanente-Fontana, Fontana, California
  - Kaiser Permanente-Fremont, Fremont, California
  - Palo Alto Medical Foundation-Fremont, Fremont, California
  - Valley Medical Oncology Consultants-Fremont, Fremont, California
  - Washington Hospital, Fremont, California
  - Kaiser Permanente-Fresno, Fresno, California
  - Kaiser Permanente South Bay, Harbor City, California
  - Kaiser Permanente-Irvine, Irvine, California
  - UC San Diego Moores Cancer Center, La Jolla, California
  - Loma Linda University Medical Center, Loma Linda, California
  - Long Beach Memorial Medical Center-Todd Cancer Institute, Long Beach, California
  - Kaiser Permanente Los Angeles Medical Center, Los Angeles, California
  - Los Angeles General Medical Center, Los Angeles, California
  - USC / Norris Comprehensive Cancer Center, Los Angeles, California
  - Kaiser Permanente West Los Angeles, Los Angeles, California
  - Cedars Sinai Medical Center, Los Angeles, California
  - Contra Costa Regional Medical Center, Martinez, California
  - Fremont - Rideout Cancer Center, Marysville, California
  - Mercy Cancer Center, Merced, California
  - Memorial Medical Center, Modesto, California
  - Kaiser Permanente-Modesto, Modesto, California
  - El Camino Hospital, Mountain View, California
  - Palo Alto Medical Foundation-Camino Division, Mountain View, California
  - Palo Alto Medical Foundation-Gynecologic Oncology, Mountain View, California
  - Northridge Hospital Medical Center, Northridge, California
  - Sutter Cancer Research Consortium, Novato, California
  - Wilma Chan Highland Hospital, Oakland, California
  - Alta Bates Summit Medical Center - Summit Campus, Oakland, California
  - Bay Area Tumor Institute, Oakland, California
  - Hematology and Oncology Associates-Oakland, Oakland, California
  - Tom K Lee Inc, Oakland, California
  - Kaiser Permanente-Oakland, Oakland, California
  - Saint Joseph Hospital - Orange, Orange, California
  - UC Irvine Health/Chao Family Comprehensive Cancer Center, Orange, California
  - Desert Regional Medical Center, Palm Springs, California
  - Palo Alto Medical Foundation Health Care, Palo Alto, California
  - Stanford Cancer Institute Palo Alto, Palo Alto, California
  - Kaiser Permanente - Panorama City, Panorama City, California
  - Keck Medical Center of USC Pasadena, Pasadena, California
  - East Bay Medical Oncology Hematology Medical Associates Inc-Pleasant Hill, Pleasant Hill, California
  - John Muir Health Cancer Medical Group, Pleasant Hill, California
  - Valley Medical Oncology Consultants, Pleasanton, California
  - Pomona Valley Hospital Medical Center, Pomona, California
  - Kaiser Permanente-Redwood City, Redwood City, California
  - Kaiser Permanente-Richmond, Richmond, California
  - Kaiser Permanente-Riverside, Riverside, California
  - Kaiser Permanente-Roseville, Roseville, California
  - Sutter Cancer Centers Radiation Oncology Services-Roseville, Roseville, California
  - Sutter Roseville Medical Center, Roseville, California
  - Sutter Medical Center Sacramento, Sacramento, California
  - University of California Davis Comprehensive Cancer Center, Sacramento, California
  - Kaiser Permanente-South Sacramento, Sacramento, California
  - Kaiser Permanente Sacramento Medical Center, Sacramento, California
  - Salinas Valley Memorial, Salinas, California
  - Kaiser Permanente-San Diego Mission, San Diego, California
  - Kaiser Permanente-San Diego Zion, San Diego, California
  - Sharp Memorial Hospital, San Diego, California
  - California Pacific Medical Center-Pacific Campus, San Francisco, California
  - Kaiser Permanente-San Francisco, San Francisco, California
  - Kaiser Permanente-Santa Teresa-San Jose, San Jose, California
  - Kaiser Permanente San Leandro, San Leandro, California
  - East Bay Medical Oncology Hematology Associates Inc, San Leandro, California
  - Kaiser Permanente-San Marcos, San Marcos, California
  - Doctors Medical Center- JC Robinson Regional Cancer Center, San Pablo, California
  - Kaiser Permanente-San Rafael, San Rafael, California
  - Kaiser Permanente Medical Center - Santa Clara, Santa Clara, California
  - Palo Alto Medical Foundation-Santa Cruz, Santa Cruz, California
  - Kaiser Permanente-Santa Rosa, Santa Rosa, California
  - Sutter Pacific Medical Foundation, Santa Rosa, California
  - Kaiser Permanente-South San Francisco, South San Francisco, California
  - Kaiser Permanente-Stockton, Stockton, California
  - Palo Alto Medical Foundation-Sunnyvale, Sunnyvale, California
  - Olive View-University of California Los Angeles Medical Center, Sylmar, California
  - Northbay Cancer Center, Vacaville, California
  - Kaiser Permanente Medical Center-Vacaville, Vacaville, California
  - Kaiser Permanente-Vallejo, Vallejo, California
  - Sutter Solano Medical Center/Cancer Center, Vallejo, California
  - Kaiser Permanente-Walnut Creek, Walnut Creek, California
  - John Muir Medical Center-Walnut Creek, Walnut Creek, California
  - Presbyterian Intercommunity Hospital, Whittier, California
  - Kaiser Permanente-Woodland Hills, Woodland Hills, California
  - San Luis Valley Regional Medical Center, Alamosa, Colorado
  - Rocky Mountain Cancer Centers-Aurora, Aurora, Colorado
  - The Medical Center of Aurora, Aurora, Colorado
  - Rocky Mountain Regional VA Medical Center, Aurora, Colorado
  - UCHealth University of Colorado Hospital, Aurora, Colorado
  - Boulder Community Foothills Hospital, Boulder, Colorado
  - Rocky Mountain Cancer Centers-Boulder, Boulder, Colorado
  - Penrose-Saint Francis Healthcare, Colorado Springs, Colorado
  - Rocky Mountain Cancer Centers-Penrose, Colorado Springs, Colorado
  - UCHealth Memorial Hospital Central, Colorado Springs, Colorado
  - Kaiser Permanente-Franklin, Denver, Colorado
  - AdventHealth Porter, Denver, Colorado
  - Colorado Blood Cancer Institute, Denver, Colorado
  - Presbyterian - Saint Lukes Medical Center - Health One, Denver, Colorado
  - Rocky Mountain Cancer Centers-Midtown, Denver, Colorado
  - Saint Joseph Hospital - Cancer Centers of Colorado, Denver, Colorado
  - Rocky Mountain Cancer Centers-Rose, Denver, Colorado
  - Rose Medical Center, Denver, Colorado
  - Western States Cancer Research NCORP, Denver, Colorado
  - CommonSpirit Cancer Center Mercy, Durango, Colorado
  - Mercy Medical Center, Durango, Colorado
  - Shaw Cancer Center, Edwards, Colorado
  - Mountain Blue Cancer Care Center - Swedish, Englewood, Colorado
  - Swedish Medical Center, Englewood, Colorado
  - Poudre Valley Hospital, Fort Collins, Colorado
  - Valley View Hospital Cancer Center, Glenwood Springs, Colorado
  - Mountain Blue Cancer Care Center, Golden, Colorado
  - Saint Mary's Hospital and Regional Medical Center, Grand Junction, Colorado
  - Banner North Colorado Medical Center, Greeley, Colorado
  - Rocky Mountain Cancer Centers-Greenwood Village, Greenwood Village, Colorado
  - Kaiser Permanente-Rock Creek, Lafayette, Colorado
  - Rocky Mountain Cancer Centers-Lakewood, Lakewood, Colorado
  - Saint Anthony Hospital, Lakewood, Colorado
  - Rocky Mountain Cancer Centers-Littleton, Littleton, Colorado
  - AdventHealth Littleton, Littleton, Colorado
  - Kaiser Permanente-Lone Tree, Lone Tree, Colorado
  - Rocky Mountain Cancer Centers-Sky Ridge, Lone Tree, Colorado
  - Sky Ridge Medical Center, Lone Tree, Colorado
  - Longmont United Hospital, Longmont, Colorado
  - Rocky Mountain Cancer Centers-Longmont, Longmont, Colorado
  - Banner North Colorado Medical Center - Loveland Campus, Loveland, Colorado
  - Montrose Memorial Hospital, Montrose, Colorado
  - AdventHealth Parker, Parker, Colorado
  - Rocky Mountain Cancer Centers-Parker, Parker, Colorado
  - Saint Mary Corwin Medical Center, Pueblo, Colorado
  - Rocky Mountain Cancer Centers - Pueblo, Pueblo, Colorado
  - North Suburban Medical Center, Thornton, Colorado
  - Rocky Mountain Cancer Centers-Thornton, Thornton, Colorado
  - Intermountain Health Lutheran Hospital, Wheat Ridge, Colorado
  - Bridgeport Hospital, Bridgeport, Connecticut
  - Danbury Hospital, Danbury, Connecticut
  - Smilow Cancer Hospital-Derby Care Center, Derby, Connecticut
  - Smilow Cancer Hospital Care Center-Fairfield, Fairfield, Connecticut
  - University of Connecticut, Farmington, Connecticut
  - Greenwich Hospital, Greenwich, Connecticut
  - Smilow Cancer Hospital Care Center - Guilford, Guilford, Connecticut
  - Hartford Hospital, Hartford, Connecticut
  - Smilow Cancer Hospital Care Center at Saint Francis, Hartford, Connecticut
  - Manchester Memorial Hospital, Manchester, Connecticut
  - Middlesex Hospital, Middletown, Connecticut
  - The Hospital of Central Connecticut, New Britain, Connecticut
  - Yale-New Haven Hospital Saint Raphael Campus, New Haven, Connecticut
  - Yale University, New Haven, Connecticut
  - Yale-New Haven Hospital North Haven Medical Center, North Haven, Connecticut
  - Norwalk Hospital, Norwalk, Connecticut
  - Eastern Connecticut Hematology and Oncology Associates, Norwich, Connecticut
  - Smilow Cancer Hospital-Orange Care Center, Orange, Connecticut
  - Smilow Cancer Hospital-Torrington Care Center, Torrington, Connecticut
  - Smilow Cancer Hospital Care Center-Trumbull, Trumbull, Connecticut
  - Harold Leever Regional Cancer Center, Waterbury, Connecticut
  - Smilow Cancer Hospital-Waterbury Care Center, Waterbury, Connecticut
  - Smilow Cancer Hospital Care Center - Waterford, Waterford, Connecticut
  - Bayhealth Hospital Kent Campus, Dover, Delaware
  - Beebe Medical Center, Lewes, Delaware
  - Bayhealth Hospital Sussex Campus, Milford, Delaware
  - Delaware Clinical and Laboratory Physicians PA, Newark, Delaware
  - Helen F Graham Cancer Center, Newark, Delaware
  - Medical Oncology Hematology Consultants PA, Newark, Delaware
  - Christiana Care Health System-Christiana Hospital, Newark, Delaware
  - Beebe Health Campus, Rehoboth Beach, Delaware
  - TidalHealth Nanticoke / Allen Cancer Center, Seaford, Delaware
  - Christiana Care Health System-Wilmington Hospital, Wilmington, Delaware
  - Kaiser Permanente-Capitol Hill Medical Center, Washington D.C., District of Columbia
  - MedStar Georgetown University Hospital, Washington D.C., District of Columbia
  - MedStar Washington Hospital Center, Washington D.C., District of Columbia
  - Sibley Memorial Hospital, Washington D.C., District of Columbia
  - George Washington University Medical Center, Washington D.C., District of Columbia
  - Mount Sinai Comprehensive Cancer Center at Aventura, Aventura, Florida
  - Boca Raton Regional Hospital, Boca Raton, Florida
  - Morton Plant Hospital, Clearwater, Florida
  - Halifax Health Medical Center-Centers for Oncology, Daytona Beach, Florida
  - AdventHealth Daytona Beach, Daytona Beach, Florida
  - Broward Health North, Deerfield Beach, Florida
  - Holy Cross Hospital, Fort Lauderdale, Florida
  - UF Health Cancer Institute - Gainesville, Gainesville, Florida
  - Saint Vincent's Medical Center, Jacksonville, Florida
  - Baptist MD Anderson Cancer Center, Jacksonville, Florida
  - Mayo Clinic in Florida, Jacksonville, Florida
  - Jupiter Medical Center, Jupiter, Florida
  - The Watson Clinic, Lakeland, Florida
  - University of Miami Miller School of Medicine-Sylvester Cancer Center, Miami, Florida
  - Advanced Medical Specialties -North, Miami, Florida
  - Miami Cancer Institute, Miami, Florida
  - Mount Sinai Medical Center, Miami Beach, Florida
  - Orlando Health Cancer Institute, Orlando, Florida
  - Sacred Heart Hospital, Pensacola, Florida
  - Saint Joseph's Hospital/Children's Hospital-Tampa, Tampa, Florida
  - Space Coast Cancer Centers-Titusville, Titusville, Florida
  - Cleveland Clinic-Weston, Weston, Florida
  - Phoebe Putney Memorial Hospital, Albany, Georgia
  - Grady Health System, Atlanta, Georgia
  - Emory University Hospital Midtown, Atlanta, Georgia
  - Piedmont Hospital, Atlanta, Georgia
  - Emory University Hospital/Winship Cancer Institute, Atlanta, Georgia
  - Atlanta Regional CCOP, Atlanta, Georgia
  - Emory Saint Joseph's Hospital, Atlanta, Georgia
  - Northside Hospital, Atlanta, Georgia
  - Augusta University Medical Center, Augusta, Georgia
  - WellStar Cobb Hospital, Austell, Georgia
  - John B Amos Cancer Center, Columbus, Georgia
  - Northside Hospital-Forsyth, Cumming, Georgia
  - Emory Decatur Hospital, Decatur, Georgia
  - Dublin Hematology Oncology Care PC, Dublin, Georgia
  - Piedmont Fayette Hospital, Fayetteville, Georgia
  - Northeast Georgia Medical Center-Gainesville, Gainesville, Georgia
  - Northside Hospital - Gwinnett, Lawrenceville, Georgia
  - Atrium Health Navicent, Macon, Georgia
  - Wellstar Kennestone Hospital, Marietta, Georgia
  - Southern Regional Medical Center, Riverdale, Georgia
  - Harbin Clinic Medical Oncology and Clinical Research, Rome, Georgia
  - Low Country Cancer Care, Savannah, Georgia
  - Memorial Health University Medical Center, Savannah, Georgia
  - Summit Cancer Care-Memorial, Savannah, Georgia
  - Lewis Cancer and Research Pavilion at Saint Joseph's/Candler, Savannah, Georgia
  - South Georgia Medical Center/Pearlman Cancer Center, Valdosta, Georgia
  - Hawaii Cancer Care Inc - Waterfront Plaza, Honolulu, Hawaii
  - Queen's Medical Center, Honolulu, Hawaii
  - Straub Clinic and Hospital, Honolulu, Hawaii
  - University of Hawaii Cancer Center, Honolulu, Hawaii
  - Queen's Cancer Center - Kuakini, Honolulu, Hawaii
  - The Cancer Center of Hawaii-Liliha, Honolulu, Hawaii
  - Kaiser Permanente Moanalua Medical Center, Honolulu, Hawaii
  - Kapiolani Medical Center for Women and Children, Honolulu, Hawaii
  - Tripler Army Medical Center, Honolulu, Hawaii
  - Castle Medical Center, Kailua, Hawaii
  - Wilcox Memorial Hospital and Kauai Medical Clinic, Lihue, Hawaii
  - Maui Memorial Medical Center, Wailuku, Hawaii
  - Pacific Cancer Institute of Maui, Wailuku, Hawaii
  - Pali Momi Medical Center, ‘Aiea, Hawaii
  - Queen's Cancer Center - Pearlridge, ‘Aiea, Hawaii
  - Saint Alphonsus Cancer Care Center-Boise, Boise, Idaho
  - Saint Luke's Cancer Institute - Boise, Boise, Idaho
  - Saint Alphonsus Cancer Care Center-Caldwell, Caldwell, Idaho
  - Kootenai Health - Coeur d'Alene, Coeur d'Alene, Idaho
  - Walter Knox Memorial Hospital, Emmett, Idaho
  - Saint Luke's Cancer Institute - Fruitland, Fruitland, Idaho
  - Saint Joseph Regional Medical Center, Lewiston, Idaho
  - Idaho Urologic Institute-Meridian, Meridian, Idaho
  - Saint Luke's Cancer Institute - Meridian, Meridian, Idaho
  - Saint Alphonsus Cancer Care Center-Nampa, Nampa, Idaho
  - Saint Luke's Cancer Institute - Nampa, Nampa, Idaho
  - Kootenai Clinic Cancer Services - Post Falls, Post Falls, Idaho
  - Kootenai Clinic Cancer Services - Sandpoint, Sandpoint, Idaho
  - Saint Luke's Cancer Institute - Twin Falls, Twin Falls, Idaho
  - OSF Saint Anthony's Health Center, Alton, Illinois
  - Rush-Copley Medical Center, Aurora, Illinois
  - Mac Neal Hospital, Berwyn, Illinois
  - OSF Saint Joseph Medical Center, Bloomington, Illinois
  - Illinois CancerCare-Bloomington, Bloomington, Illinois
  - Graham Hospital Association, Canton, Illinois
  - Illinois CancerCare-Canton, Canton, Illinois
  - Memorial Hospital of Carbondale, Carbondale, Illinois
  - Illinois CancerCare-Carthage, Carthage, Illinois
  - Memorial Hospital, Carthage, Illinois
  - Centralia Oncology Clinic, Centralia, Illinois
  - Mount Sinai Hospital Medical Center, Chicago, Illinois
  - Hematology and Oncology Associates, Chicago, Illinois
  - Northwestern University, Chicago, Illinois
  - John H Stroger Jr Hospital of Cook County, Chicago, Illinois
  - University of Illinois, Chicago, Illinois
  - Presence Resurrection Medical Center, Chicago, Illinois
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - Weiss Memorial Hospital, Chicago, Illinois
  - Carle at The Riverfront, Danville, Illinois
  - Cancer Care Specialists of Illinois - Decatur, Decatur, Illinois
  - Decatur Memorial Hospital, Decatur, Illinois
  - Heartland Cancer Research NCORP, Decatur, Illinois
  - Northwestern Medicine Cancer Center Kishwaukee, DeKalb, Illinois
  - Advocate Good Samaritan Hospital, Downers Grove, Illinois
  - Carle Physician Group-Effingham, Effingham, Illinois
  - Crossroads Cancer Center, Effingham, Illinois
  - Advocate Sherman Hospital, Elgin, Illinois
  - Elmhurst Memorial Hospital, Elmhurst, Illinois
  - Eureka Hospital, Eureka, Illinois
  - Illinois CancerCare-Eureka, Eureka, Illinois
  - Saint Francis Hospital, Evanston, Illinois
  - Freeport Memorial Hospital/Leonard C Ferguson Cancer Center, Freeport, Illinois
  - Illinois CancerCare-Galesburg, Galesburg, Illinois
  - Western Illinois Cancer Treatment Center, Galesburg, Illinois
  - Ingalls Memorial Hospital, Harvey, Illinois
  - Illinois CancerCare-Havana, Havana, Illinois
  - Mason District Hospital, Havana, Illinois
  - Hematology Oncology Associates of Illinois-Highland Park, Highland Park, Illinois
  - Hinsdale Hematology Oncology Associates Incorporated, Hinsdale, Illinois
  - UChicago Medicine AdventHealth Cancer Institute Hinsdale, Hinsdale, Illinois
  - Presence Saint Mary's Hospital, Kankakee, Illinois
  - Illinois CancerCare-Kewanee Clinic, Kewanee, Illinois
  - AMITA Health Adventist Medical Center, La Grange, Illinois
  - AMG Libertyville - Oncology, Libertyville, Illinois
  - Illinois CancerCare-Macomb, Macomb, Illinois
  - Mcdonough District Hospital, Macomb, Illinois
  - Carle Physician Group-Mattoon/Charleston, Mattoon, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - Garneau, Stewart C MD (UIA Investigator), Moline, Illinois
  - Porubcin, Michael MD (UIA Investigator), Moline, Illinois
  - Spector, David MD (UIA Investigator), Moline, Illinois
  - Trinity Medical Center, Moline, Illinois
  - Holy Family Medical Center, Monmouth, Illinois
  - Illinois CancerCare-Monmouth, Monmouth, Illinois
  - SSM Health Good Samaritan, Mount Vernon, Illinois
  - Edward Hospital/Cancer Center, Naperville, Illinois
  - UC Comprehensive Cancer Center at Silver Cross, New Lenox, Illinois
  - Illinois Cancer Specialists-Niles, Niles, Illinois
  - Carle BroMenn Medical Center, Normal, Illinois
  - Carle Cancer Institute Normal, Normal, Illinois
  - Illinois CancerCare-Community Cancer Center, Normal, Illinois
  - Mid-Illinois Hematology Oncology Associates Limited, Normal, Illinois
  - Cancer Care Center of O'Fallon, O'Fallon, Illinois
  - Advocate Christ Medical Center, Oak Lawn, Illinois
  - Illinois CancerCare-Ottawa Clinic, Ottawa, Illinois
  - Ottawa Regional Hospital and Healthcare Center, Ottawa, Illinois
  - Radiation Oncology of Northern Illinois, Ottawa, Illinois
  - Advocate Lutheran General Hospital, Park Ridge, Illinois
  - Illinois CancerCare-Pekin, Pekin, Illinois
  - OSF Saint Francis Radiation Oncology at Pekin, Pekin, Illinois
  - Proctor Hospital, Peoria, Illinois
  - Illinois CancerCare-Peoria, Peoria, Illinois
  - OSF Saint Francis Radiation Oncology at Peoria Cancer Center, Peoria, Illinois
  - Methodist Medical Center of Illinois, Peoria, Illinois
  - OSF Saint Francis Medical Center, Peoria, Illinois
  - Illinois CancerCare-Peru, Peru, Illinois
  - Illinois Valley Hospital, Peru, Illinois
  - Valley Radiation Oncology, Peru, Illinois
  - Illinois CancerCare-Princeton, Princeton, Illinois
  - Perry Memorial Hospital, Princeton, Illinois
  - West Suburban Medical Center, River Forest, Illinois
  - Swedish American Hospital, Rockford, Illinois
  - UW Health Carbone Cancer Center Rockford, Rockford, Illinois
  - Hematology Oncology Associates of Illinois - Skokie, Skokie, Illinois
  - Illinois CancerCare-Spring Valley, Spring Valley, Illinois
  - Central Illinois Hematology Oncology Center, Springfield, Illinois
  - Southern Illinois University School of Medicine, Springfield, Illinois
  - Springfield Clinic, Springfield, Illinois
  - Springfield Memorial Hospital, Springfield, Illinois
  - Carle Cancer Center, Urbana, Illinois
  - The Carle Foundation Hospital, Urbana, Illinois
  - Rush-Copley Healthcare Center, Yorkville, Illinois
  - Franciscan Saint Francis Health-Beech Grove, Beech Grove, Indiana
  - IU Health North Hospital, Carmel, Indiana
  - Michiana Hematology Oncology PC-Crown Point, Crown Point, Indiana
  - Elkhart Clinic, Elkhart, Indiana
  - Michiana Hematology Oncology PC-Elkhart, Elkhart, Indiana
  - Elkhart General Hospital, Elkhart, Indiana
  - Deaconess Clinic Downtown, Evansville, Indiana
  - Fort Wayne Medical Oncology and Hematology Inc-Parkview, Fort Wayne, Indiana
  - Indiana University/Melvin and Bren Simon Cancer Center, Indianapolis, Indiana
  - IU Health Methodist Hospital, Indianapolis, Indiana
  - Sidney and Lois Eskenazi Hospital, Indianapolis, Indiana
  - IU Health Central Indiana Cancer Centers-East, Indianapolis, Indiana
  - Franciscan Health Indianapolis, Indianapolis, Indiana
  - Springmill Medical Center, Indianapolis, Indiana
  - Community Howard Regional Health, Kokomo, Indiana
  - IU Health La Porte Hospital, La Porte, Indiana
  - IU Health Arnett Cancer Care, Lafayette, Indiana
  - Premier Oncology Hematology Associates, Merrillville, Indiana
  - Franciscan Saint Anthony Health-Michigan City, Michigan City, Indiana
  - Woodland Cancer Care Center, Michigan City, Indiana
  - Memorial Regional Cancer Center Day Road, Mishawaka, Indiana
  - Michiana Hematology Oncology PC-Mishawaka, Mishawaka, Indiana
  - Saint Joseph Regional Medical Center-Mishawaka, Mishawaka, Indiana
  - IU Health Ball Memorial Hospital, Muncie, Indiana
  - Chancellor Center for Oncology, Newburgh, Indiana
  - Michiana Hematology Oncology PC-Plymouth, Plymouth, Indiana
  - Reid Health, Richmond, Indiana
  - Memorial Hospital of South Bend, South Bend, Indiana
  - South Bend Clinic, South Bend, Indiana
  - Northern Indiana Cancer Research Consortium, South Bend, Indiana
  - Porter Memorial Hospital, Valparaiso, Indiana
  - Michiana Hematology Oncology PC-Westville, Westville, Indiana
  - Mary Greeley Medical Center, Ames, Iowa
  - McFarland Clinic - Ames, Ames, Iowa
  - Constantinou, Costas L MD (UIA Investigator), Bettendorf, Iowa
  - McFarland Clinic - Boone, Boone, Iowa
  - Physicians' Clinic of Iowa PC, Cedar Rapids, Iowa
  - Saint Luke's Hospital, Cedar Rapids, Iowa
  - Mercy Hospital, Cedar Rapids, Iowa
  - Oncology Associates at Mercy Medical Center, Cedar Rapids, Iowa
  - Mercy Cancer Center-West Lakes, Clive, Iowa
  - UI Health Care Mission Cancer and Blood - West Des Moines Clinic, Clive, Iowa
  - Alegent Health Mercy Hospital, Council Bluffs, Iowa
  - Heartland Oncology and Hematology LLP, Council Bluffs, Iowa
  - Greater Regional Medical Center, Creston, Iowa
  - MercyOne Genesis Davenport Medical Center, Davenport, Iowa
  - Iowa Methodist Medical Center, Des Moines, Iowa
  - UI Health Care Mission Cancer and Blood - Des Moines Clinic, Des Moines, Iowa
  - Mercy Medical Center - Des Moines, Des Moines, Iowa
  - UI Health Care Mission Cancer and Blood - Laurel Clinic, Des Moines, Iowa
  - Iowa Lutheran Hospital, Des Moines, Iowa
  - JCHC McCreery Cancer Center, Fairfield, Iowa
  - McFarland Clinic - Trinity Cancer Center, Fort Dodge, Iowa
  - McFarland Clinic - Jefferson, Jefferson, Iowa
  - McFarland Clinic - Marshalltown, Marshalltown, Iowa
  - Mercy Medical Center - North Iowa, Mason City, Iowa
  - Ottumwa Regional Health Center, Ottumwa, Iowa
  - Siouxland Regional Cancer Center, Sioux City, Iowa
  - Mercy Medical Center-Sioux City, Sioux City, Iowa
  - Saint Luke's Regional Medical Center, Sioux City, Iowa
  - MercyOne Waterloo Cancer Center, Waterloo, Iowa
  - Methodist West Hospital, West Des Moines, Iowa
  - Mercy Medical Center-West Lakes, West Des Moines, Iowa
  - Cancer Center of Kansas - Chanute, Chanute, Kansas
  - Cancer Center of Kansas - Dodge City, Dodge City, Kansas
  - Cancer Center of Kansas - El Dorado, El Dorado, Kansas
  - Newman Regional Health, Emporia, Kansas
  - Cancer Center of Kansas - Fort Scott, Fort Scott, Kansas
  - Saint Catherine Hospital, Garden City, Kansas
  - Saint Rose Ambulatory and Surgery Center, Great Bend, Kansas
  - HaysMed, Hays, Kansas
  - Hutchinson Regional Medical Center, Hutchinson, Kansas
  - Cancer Center of Kansas-Independence, Independence, Kansas
  - Providence Medical Center, Kansas City, Kansas
  - University of Kansas Cancer Center-West, Kansas City, Kansas
  - University of Kansas Cancer Center, Kansas City, Kansas
  - Cancer Center of Kansas-Kingman, Kingman, Kansas
  - Lawrence Memorial Hospital, Lawrence, Kansas
  - Kansas Institute of Medicine Cancer and Blood Center, Lenexa, Kansas
  - Minimally Invasive Surgery Hospital, Lenexa, Kansas
  - Cancer Center of Kansas-Liberal, Liberal, Kansas
  - Cancer Center of Kansas-Manhattan, Manhattan, Kansas
  - Cancer Center of Kansas - McPherson, McPherson, Kansas
  - Cancer Center of Kansas - Newton, Newton, Kansas
  - The University of Kansas Cancer Center - Olathe, Olathe, Kansas
  - Menorah Medical Center, Overland Park, Kansas
  - University of Kansas Cancer Center-Overland Park, Overland Park, Kansas
  - Saint Luke's South Hospital, Overland Park, Kansas
  - Cancer Center of Kansas - Parsons, Parsons, Kansas
  - Mercy Hospital Pittsburg, Pittsburg, Kansas
  - Kansas City NCI Community Oncology Research Program, Prairie Village, Kansas
  - Cancer Center of Kansas - Pratt, Pratt, Kansas
  - Cancer Center of Kansas - Salina, Salina, Kansas
  - Salina Regional Health Center, Salina, Kansas
  - Cotton O'Neil Cancer Center / Stormont Vail Health, Topeka, Kansas
  - University of Kansas Health System Saint Francis Campus, Topeka, Kansas
  - Cancer Center of Kansas - Wellington, Wellington, Kansas
  - Associates In Womens Health, Wichita, Kansas
  - Cancer Center of Kansas-Wichita Medical Arts Tower, Wichita, Kansas
  - Ascension Via Christi Hospitals Wichita, Wichita, Kansas
  - Cancer Center of Kansas - Wichita, Wichita, Kansas
  - Wesley Medical Center, Wichita, Kansas
  - Wichita NCI Community Oncology Research Program, Wichita, Kansas
  - Cancer Center of Kansas - Winfield, Winfield, Kansas
  - King's Daughter's Medical Center, Ashland, Kentucky
  - Flaget Memorial Hospital, Bardstown, Kentucky
  - Baptist Health Corbin, Corbin, Kentucky
  - Commonwealth Cancer Center-Corbin, Corbin, Kentucky
  - Oncology Hematology Care Inc-Crestview, Crestview Hills, Kentucky
  - Saint Elizabeth Healthcare Edgewood, Edgewood, Kentucky
  - Baptist Health Hardin, Elizabethtown, Kentucky
  - Saint Elizabeth Healthcare Fort Thomas, Fort Thomas, Kentucky
  - Baptist Health Lexington, Lexington, Kentucky
  - Saint Joseph Radiation Oncology Resource Center, Lexington, Kentucky
  - Saint Joseph Hospital East, Lexington, Kentucky
  - University of Kentucky/Markey Cancer Center, Lexington, Kentucky
  - Saint Joseph London, London, Kentucky
  - Jewish Hospital, Louisville, Kentucky
  - The James Graham Brown Cancer Center at University of Louisville, Louisville, Kentucky
  - Saints Mary and Elizabeth Hospital, Louisville, Kentucky
  - UofL Health Medical Center Northeast, Louisville, Kentucky
  - Baptist Health Madisonville/Merle Mahr Cancer Center, Madisonville, Kentucky
  - Owensboro Health Mitchell Memorial Cancer Center, Owensboro, Kentucky
  - Baptist Health Paducah, Paducah, Kentucky
  - Jewish Hospital Medical Center South, Shepherdsville, Kentucky
  - Christus Saint Frances Cabrini Hospital, Alexandria, Louisiana
  - LSU Health Baton Rouge-North Clinic, Baton Rouge, Louisiana
  - Baton Rouge General Medical Center, Baton Rouge, Louisiana
  - Our Lady of the Lake Physician Group, Baton Rouge, Louisiana
  - Hematology/Oncology Clinic PLLC, Baton Rouge, Louisiana
  - Louisiana Hematology Oncology Associates LLC, Baton Rouge, Louisiana
  - Mary Bird Perkins Cancer Center, Baton Rouge, Louisiana
  - Ochsner Health Center-Summa, Baton Rouge, Louisiana
  - Mary Bird Perkins Cancer Center - Covington, Covington, Louisiana
  - Ochsner Health Center-Covington, Covington, Louisiana
  - Mary Bird Perkins Cancer Center - Houma, Houma, Louisiana
  - Ochsner Medical Center Kenner, Kenner, Louisiana
  - West Jefferson Medical Center, Marrero, Louisiana
  - East Jefferson General Hospital, Metairie, Louisiana
  - Robert Veith MD LLC, Metairie, Louisiana
  - Ochsner LSU Health Monroe Medical Center, Monroe, Louisiana
  - Louisiana State University Health Science Center, New Orleans, Louisiana
  - Tulane University School of Medicine, New Orleans, Louisiana
  - University Medical Center New Orleans, New Orleans, Louisiana
  - Ochsner Baptist Medical Center, New Orleans, Louisiana
  - Ochsner Medical Center Jefferson, New Orleans, Louisiana
  - LSU Health Sciences Center at Shreveport, Shreveport, Louisiana
  - Highland Clinic, Shreveport, Louisiana
  - Harold Alfond Center for Cancer Care, Augusta, Maine
  - Eastern Maine Medical Center, Bangor, Maine
  - Lafayette Family Cancer Center-EMMC, Brewer, Maine
  - Mercy Hospital, Portland, Maine
  - Penobscot Bay Medical Center, Rockport, Maine
  - New England Cancer Specialists, Westbrook, Maine
  - Mercy Medical Center, Baltimore, Maryland
  - Greater Baltimore Medical Center, Baltimore, Maryland
  - Sinai Hospital of Baltimore, Baltimore, Maryland
  - MedStar Union Memorial Hospital, Baltimore, Maryland
  - MedStar Good Samaritan Hospital, Baltimore, Maryland
  - Kaiser Permanente-Woodlawn Medical Center, Baltimore, Maryland
  - Johns Hopkins University/Sidney Kimmel Cancer Center, Baltimore, Maryland
  - Suburban Hospital, Bethesda, Maryland
  - Walter Reed National Military Medical Center, Bethesda, Maryland
  - University of Maryland Shore Medical Center at Easton, Easton, Maryland
  - Christiana Care - Union Hospital, Elkton, Maryland
  - Frederick Memorial Hospital, Frederick, Maryland
  - Kaiser Permanente-Gaithersburg Medical Center, Gaithersburg, Maryland
  - Kaiser Permanente - Kensington Medical Center, Kensington, Maryland
  - Kaiser Permanente - Largo Medical Center, Largo, Maryland
  - MedStar Montgomery Medical Center, Olney, Maryland
  - Northwest Hospital Center, Randallstown, Maryland
  - TidalHealth Peninsula Regional, Salisbury, Maryland
  - William E Kahlert Regional Cancer Center/Sinai Hospital, Westminster, Maryland
  - Sturdy Memorial Hospital, Attleboro, Massachusetts
  - Beverly Hospital, Beverly, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Dana-Farber Cancer Institute at Boston Medical Center - Brighton, Brighton, Massachusetts
  - Lahey Hospital and Medical Center, Burlington, Massachusetts
  - Mass General/North Shore Cancer Center, Danvers, Massachusetts
  - Saint Anne's Hospital, Fall River, Massachusetts
  - Addison Gilbert Hospital, Gloucester, Massachusetts
  - Cape Cod Hospital, Hyannis, Massachusetts
  - Lowell General Hospital, Lowell, Massachusetts
  - Holy Family Hospital, Methuen, Massachusetts
  - Dana-Farber/Brigham and Women's Cancer Center at Milford Regional, Milford, Massachusetts
  - Newton-Wellesley Hospital, Newton, Massachusetts
  - Berkshire Medical Center - Cancer Center, Pittsfield, Massachusetts
  - Beth Israel Deaconess Hospital-Plymouth, Plymouth, Massachusetts
  - Dana Farber Community Cancer Care-Quincy, Quincy, Massachusetts
  - Dana-Farber/Brigham and Women's Cancer Center at South Shore, South Weymouth, Massachusetts
  - UMass Memorial Medical Center - University Campus, Worcester, Massachusetts
  - Bixby Medical Center, Adrian, Michigan
  - Hickman Cancer Center, Adrian, Michigan
  - Michigan Cancer Research Consortium NCORP, Ann Arbor, Michigan
  - Trinity Health Saint Joseph Mercy Hospital Ann Arbor, Ann Arbor, Michigan
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Bronson Battle Creek, Battle Creek, Michigan
  - McLaren Cancer Institute-Bay City, Bay City, Michigan
  - Spectrum Health Big Rapids Hospital, Big Rapids, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology - Brighton, Brighton, Michigan
  - Trinity Health Medical Center - Brighton, Brighton, Michigan
  - Henry Ford Cancer Institute-Downriver, Brownstown, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology - Canton, Canton, Michigan
  - Trinity Health Medical Center - Canton, Canton, Michigan
  - Caro Cancer Center, Caro, Michigan
  - Chelsea Hospital, Chelsea, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology - Chelsea Hospital, Chelsea, Michigan
  - Hematology Oncology Consultants-Clarkston, Clarkston, Michigan
  - McLaren Cancer Institute-Clarkston, Clarkston, Michigan
  - Newland Medical Associates-Clarkston, Clarkston, Michigan
  - Henry Ford Macomb Hospital-Clinton Township, Clinton Township, Michigan
  - Huron Valley-Sinai Hospital, Commerce, Michigan
  - Corewell Health Dearborn Hospital, Dearborn, Michigan
  - Henry Ford Medical Center-Fairlane, Dearborn, Michigan
  - Wayne State University/Karmanos Cancer Institute, Detroit, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - Henry Ford Health Saint John Hospital, Detroit, Michigan
  - Henry Ford River District Hospital, East China Township, Michigan
  - OSF Saint Francis Hospital and Medical Group, Escanaba, Michigan
  - Weisberg Cancer Treatment Center, Farmington Hills, Michigan
  - Corewell Health Farmington Hills Hospital, Farmington Hills, Michigan
  - Cancer Hematology Centers - Flint, Flint, Michigan
  - Genesee Hematology Oncology PC, Flint, Michigan
  - Genesys Hurley Cancer Institute, Flint, Michigan
  - Hurley Medical Center, Flint, Michigan
  - Genesys Regional Medical Center-West Flint Campus, Flint, Michigan
  - McLaren Cancer Institute-Flint, Flint, Michigan
  - Singh and Arora Hematology Oncology PC, Flint, Michigan
  - Cancer Research Consortium of West Michigan NCORP, Grand Rapids, Michigan
  - Corewell Health Grand Rapids Hospitals - Butterworth Hospital, Grand Rapids, Michigan
  - Trinity Health Grand Rapids Hospital, Grand Rapids, Michigan
  - Henry Ford Saint John Hospital - Academic, Grosse Pointe Woods, Michigan
  - Henry Ford Saint John Hospital - Breast, Grosse Pointe Woods, Michigan
  - Henry Ford Saint John Hospital - Van Elslander, Grosse Pointe Woods, Michigan
  - Allegiance Health, Jackson, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - Beacon Kalamazoo, Kalamazoo, Michigan
  - Karmanos Cancer Institute at McLaren Greater Lansing, Lansing, Michigan
  - University of Michigan Health - Sparrow Lansing, Lansing, Michigan
  - McLaren Cancer Institute-Lapeer Region, Lapeer, Michigan
  - Hope Cancer Clinic, Livonia, Michigan
  - Trinity Health Saint Mary Mercy Livonia Hospital, Livonia, Michigan
  - Henry Ford Saint John Hospital - Macomb Medical, Macomb, Michigan
  - Henry Ford Warren Hospital - Breast Macomb, Macomb, Michigan
  - Saint Mary's Oncology/Hematology Associates of Marlette, Marlette, Michigan
  - UP Health System Marquette, Marquette, Michigan
  - MyMichigan Medical Center Midland, Midland, Michigan
  - Mercy Memorial Hospital, Monroe, Michigan
  - Monroe Cancer Center, Monroe, Michigan
  - Toledo Clinic Cancer Centers-Monroe, Monroe, Michigan
  - McLaren Cancer Institute-Macomb, Mount Clemens, Michigan
  - McLaren Cancer Institute-Central Michigan, Mount Pleasant, Michigan
  - Trinity Health Muskegon Hospital, Muskegon, Michigan
  - Corewell Health Lakeland Hospitals - Niles Hospital, Niles, Michigan
  - Henry Ford Health Providence Novi Hospital, Novi, Michigan
  - Henry Ford Medical Center-Columbus, Novi, Michigan
  - McLaren Cancer Institute-Northern Michigan, Petoskey, Michigan
  - Hope Cancer Center, Pontiac, Michigan
  - Michigan Healthcare Professionals Pontiac, Pontiac, Michigan
  - Newland Medical Associates-Pontiac, Pontiac, Michigan
  - Trinity Health Saint Joseph Mercy Oakland Hospital, Pontiac, Michigan
  - Lake Huron Medical Center, Port Huron, Michigan
  - Corewell Health Reed City Hospital, Reed City, Michigan
  - Henry Ford Rochester Hospital, Rochester Hills, Michigan
  - Corewell Health William Beaumont University Hospital, Royal Oak, Michigan
  - MyMichigan Medical Center Saginaw, Saginaw, Michigan
  - Oncology Hematology Associates of Saginaw Valley PC, Saginaw, Michigan
  - Corewell Health Lakeland Hospitals - Marie Yeager Cancer Center, Saint Joseph, Michigan
  - Corewell Health Lakeland Hospitals - Saint Joseph Hospital, Saint Joseph, Michigan
  - Henry Ford Health Providence Southfield Hospital, Southfield, Michigan
  - Bhadresh Nayak MD PC-Sterling Heights, Sterling Heights, Michigan
  - MyMichigan Medical Center Tawas, Tawas City, Michigan
  - Munson Medical Center, Traverse City, Michigan
  - Corewell Health Beaumont Troy Hospital, Troy, Michigan
  - Advanced Breast Care Center PLLC, Warren, Michigan
  - Henry Ford Health Warren Hospital, Warren, Michigan
  - Henry Ford Madison Heights Hospital - Breast, Warren, Michigan
  - Henry Ford Warren Hospital - GLCMS, Warren, Michigan
  - Macomb Hematology Oncology PC, Warren, Michigan
  - Henry Ford West Bloomfield Hospital, West Bloomfield, Michigan
  - Saint Mary's Oncology/Hematology Associates of West Branch, West Branch, Michigan
  - University of Michigan Health - West, Wyoming, Michigan
  - Huron Gastroenterology PC, Ypsilanti, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology Ann Arbor Campus, Ypsilanti, Michigan
  - Medini, Eitan MD (UIA Investigator), Alexandria, Minnesota
  - Fairview Ridges Hospital, Burnsville, Minnesota
  - Mercy Hospital, Coon Rapids, Minnesota
  - Saint Luke's Hospital of Duluth, Duluth, Minnesota
  - Fairview Southdale Hospital, Edina, Minnesota
  - Unity Hospital, Fridley, Minnesota
  - Hutchinson Area Health Care, Hutchinson, Minnesota
  - Mayo Clinic Health Systems-Mankato, Mankato, Minnesota
  - Fairview Clinics and Surgery Center Maple Grove, Maple Grove, Minnesota
  - Minnesota Oncology Hematology PA-Maplewood, Maplewood, Minnesota
  - Saint John's Hospital - Healtheast, Maplewood, Minnesota
  - Abbott-Northwestern Hospital, Minneapolis, Minnesota
  - Hennepin County Medical Center, Minneapolis, Minnesota
  - Health Partners Inc, Minneapolis, Minnesota
  - New Ulm Medical Center, New Ulm, Minnesota
  - North Memorial Medical Health Center, Robbinsdale, Minnesota
  - Mayo Clinic in Rochester, Rochester, Minnesota
  - Coborn Cancer Center at Saint Cloud Hospital, Saint Cloud, Minnesota
  - Saint Cloud Hospital, Saint Cloud, Minnesota
  - Metro Minnesota Community Oncology Research Consortium, Saint Louis Park, Minnesota
  - Park Nicollet Clinic - Saint Louis Park, Saint Louis Park, Minnesota
  - Regions Hospital, Saint Paul, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - Saint Francis Regional Medical Center, Shakopee, Minnesota
  - Lakeview Hospital, Stillwater, Minnesota
  - Ridgeview Medical Center, Waconia, Minnesota
  - Rice Memorial Hospital, Willmar, Minnesota
  - Minnesota Oncology Hematology PA-Woodbury, Woodbury, Minnesota
  - Fairview Lakes Medical Center, Wyoming, Minnesota
  - Gulfport Memorial Hospital, Gulfport, Mississippi
  - Hattiesburg Clinic - Hematology/Oncology Clinic, Hattiesburg, Mississippi
  - Forrest General Hospital / Cancer Center, Hattiesburg, Mississippi
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Singing River Hospital, Pascagoula, Mississippi
  - Central Care Cancer Center - Bolivar, Bolivar, Missouri
  - Parkland Health Center-Bonne Terre, Bonne Terre, Missouri
  - Cox Cancer Center Branson, Branson, Missouri
  - Mercy Cancer Center - Cape Girardeau, Cape Girardeau, Missouri
  - Saint Francis Medical Center, Cape Girardeau, Missouri
  - Saint Luke's Hospital, Chesterfield, Missouri
  - Siteman Cancer Center at Saint Peters Hospital, City of Saint Peters, Missouri
  - MU Health - University Hospital/Ellis Fischel Cancer Center, Columbia, Missouri
  - Siteman Cancer Center at West County Hospital, Creve Coeur, Missouri
  - Centerpoint Medical Center LLC, Independence, Missouri
  - MU Health Care Goldschmidt Cancer Center, Jefferson City, Missouri
  - Freeman Health System, Joplin, Missouri
  - Mercy Hospital Joplin, Joplin, Missouri
  - University Health Truman Medical Center, Kansas City, Missouri
  - Saint Luke's Hospital of Kansas City, Kansas City, Missouri
  - Saint Joseph Health Center, Kansas City, Missouri
  - North Kansas City Hospital, Kansas City, Missouri
  - Heartland Hematology and Oncology Associates Incorporated, Kansas City, Missouri
  - The University of Kansas Cancer Center-South, Kansas City, Missouri
  - Research Medical Center, Kansas City, Missouri
  - University of Kansas Cancer Center - North, Kansas City, Missouri
  - University of Kansas Cancer Center - Lee's Summit, Lee's Summit, Missouri
  - Saint Luke's East - Lee's Summit, Lee's Summit, Missouri
  - Liberty Hospital, Liberty, Missouri
  - Mercy Clinic-Rolla-Cancer and Hematology, Rolla, Missouri
  - Phelps Health Delbert Day Cancer Institute, Rolla, Missouri
  - Heartland Regional Medical Center, Saint Joseph, Missouri
  - Sainte Genevieve County Memorial Hospital, Sainte Genevieve, Missouri
  - Cancer Research for the Ozarks NCORP, Springfield, Missouri
  - Mercy Hospital Springfield, Springfield, Missouri
  - CoxHealth South Hospital, Springfield, Missouri
  - SSM Health Saint Louis University Hospital, St Louis, Missouri
  - Mercy Infusion Center - Chippewa, St Louis, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Missouri Baptist Medical Center, St Louis, Missouri
  - Siteman Cancer Center at Christian Hospital, St Louis, Missouri
  - Comprehensive Cancer Care PC, St Louis, Missouri
  - Mercy Hospital Saint Louis, St Louis, Missouri
  - Saint Louis-Cape Girardeau CCOP, St Louis, Missouri
  - Missouri Baptist Sullivan Hospital, Sullivan, Missouri
  - BJC Outpatient Center at Sunset Hills, Sunset Hills, Missouri
  - Community Hospital of Anaconda, Anaconda, Montana
  - Billings Clinic Cancer Center, Billings, Montana
  - Saint Vincent Healthcare, Billings, Montana
  - Montana Cancer Consortium NCORP, Billings, Montana
  - Saint Vincent Frontier Cancer Center, Billings, Montana
  - Bozeman Health Deaconess Hospital, Bozeman, Montana
  - Saint James Community Hospital and Cancer Treatment Center, Butte, Montana
  - Benefis Sletten Cancer Institute, Great Falls, Montana
  - Great Falls Clinic, Great Falls, Montana
  - Northern Montana Hospital, Havre, Montana
  - Saint Peter's Community Hospital, Helena, Montana
  - Glacier Oncology PLLC, Kalispell, Montana
  - Kalispell Medical Oncology, Kalispell, Montana
  - Logan Health Medical Center, Kalispell, Montana
  - Montana Cancer Specialists, Missoula, Montana
  - Saint Patrick Hospital - Community Hospital, Missoula, Montana
  - Community Medical Center, Missoula, Montana
  - Nebraska Cancer Specialists/Oncology Hematology West PC, Grand Island, Nebraska
  - Fred and Pamela Buffett Cancer Center - Kearney, Kearney, Nebraska
  - CHI Health Good Samaritan, Kearney, Nebraska
  - Nebraska Hematology and Oncology, Lincoln, Nebraska
  - Nebraska Cancer Research Center, Lincoln, Nebraska
  - Saint Elizabeth Regional Medical Center, Lincoln, Nebraska
  - Cancer Partners of Nebraska, Lincoln, Nebraska
  - Faith Regional Health Services Carson Cancer Center, Norfolk, Nebraska
  - Great Plains Health Callahan Cancer Center, North Platte, Nebraska
  - Missouri Valley Cancer Consortium, Omaha, Nebraska
  - Nebraska Methodist Hospital, Omaha, Nebraska
  - Alegent Health Immanuel Medical Center, Omaha, Nebraska
  - Hematology and Oncology Consultants PC, Omaha, Nebraska
  - Alegent Health Bergan Mercy Medical Center, Omaha, Nebraska
  - Nebraska Cancer Specialists - Omaha, Omaha, Nebraska
  - Alegent Health Lakeside Hospital, Omaha, Nebraska
  - Oncology Hematology West PC, Omaha, Nebraska
  - Urology Cancer Center PC, Omaha, Nebraska
  - Creighton University Medical Center, Omaha, Nebraska
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Midlands Community Hospital, Papillion, Nebraska
  - Regional West Medical Center Cancer Center, Scottsbluff, Nebraska
  - Cancer and Blood Specialists-Henderson, Henderson, Nevada
  - Comprehensive Cancer Centers of Nevada - Henderson, Henderson, Nevada
  - Comprehensive Cancer Centers of Nevada-Horizon Ridge, Henderson, Nevada
  - Las Vegas Cancer Center-Henderson, Henderson, Nevada
  - OptumCare Cancer Care at Seven Hills, Henderson, Nevada
  - Comprehensive Cancer Centers of Nevada-Southeast Henderson, Henderson, Nevada
  - Oncology Las Vegas - Henderson, Henderson, Nevada
  - Desert West Surgery, Las Vegas, Nevada
  - OptumCare Cancer Care at Charleston, Las Vegas, Nevada
  - University Medical Center of Southern Nevada, Las Vegas, Nevada
  - Cancer and Blood Specialists-Shadow, Las Vegas, Nevada
  - Radiation Oncology Centers of Nevada Central, Las Vegas, Nevada
  - HealthCare Partners Medical Group Oncology/Hematology-Maryland Parkway, Las Vegas, Nevada
  - HealthCare Partners Medical Group Oncology/Hematology-San Martin, Las Vegas, Nevada
  - Radiation Oncology Centers of Nevada Southeast, Las Vegas, Nevada
  - Nevada Cancer Research Foundation NCORP, Las Vegas, Nevada
  - Cancer Therapy and Integrative Medicine, Las Vegas, Nevada
  - Ann M Wierman MD LTD, Las Vegas, Nevada
  - Cancer and Blood Specialists-Tenaya, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada - Northwest, Las Vegas, Nevada
  - HealthCare Partners Medical Group Oncology/Hematology-Tenaya, Las Vegas, Nevada
  - Oncology Las Vegas - Tenaya, Las Vegas, Nevada
  - OptumCare Cancer Care at MountainView, Las Vegas, Nevada
  - Alliance for Childhood Diseases/Cure 4 the Kids Foundation, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada-Summerlin, Las Vegas, Nevada
  - Summerlin Hospital Medical Center, Las Vegas, Nevada
  - Las Vegas Cancer Center-Medical Center, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada, Las Vegas, Nevada
  - OptumCare Cancer Care at Fort Apache, Las Vegas, Nevada
  - HealthCare Partners Medical Group Oncology/Hematology-Centennial Hills, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada - Central Valley, Las Vegas, Nevada
  - Hope Cancer Care of Nevada-Pahrump, Pahrump, Nevada
  - Renown Regional Medical Center, Reno, Nevada
  - Saint Mary's Regional Medical Center, Reno, Nevada
  - Radiation Oncology Associates, Reno, Nevada
  - Parkland Medical Center, Derry, New Hampshire
  - Wentworth-Douglass Hospital, Dover, New Hampshire
  - Cheshire Medical Center-Dartmouth-Hitchcock Keene, Keene, New Hampshire
  - Dartmouth Hitchcock Medical Center/Dartmouth Cancer Center, Lebanon, New Hampshire
  - The Dana-Farber Cancer Institute at Londonderry, Londonderry, New Hampshire
  - Dartmouth Cancer Center - Manchester, Manchester, New Hampshire
  - Foundation Medical Partners, Nashua, New Hampshire
  - Dartmouth Cancer Center - Nashua, Nashua, New Hampshire
  - Portsmouth Regional Hospital, Portsmouth, New Hampshire
  - Memorial Sloan Kettering Basking Ridge, Basking Ridge, New Jersey
  - Cooper Hospital University Medical Center, Camden, New Jersey
  - AtlantiCare Health Park-Cape May Court House, Cape May Court House, New Jersey
  - AtlantiCare Surgery Center, Egg Harbor, New Jersey
  - Englewood Hospital and Medical Center, Englewood, New Jersey
  - Hackensack University Medical Center, Hackensack, New Jersey
  - The Cancer Institute of New Jersey Hamilton, Hamilton, New Jersey
  - Saint Barnabas Medical Center, Livingston, New Jersey
  - Monmouth Medical Center, Long Branch, New Jersey
  - Morristown Medical Center, Morristown, New Jersey
  - Virtua Memorial, Mount Holly, New Jersey
  - Inspira Medical Center Mullica Hill, Mullica Hill, New Jersey
  - Saint Peter's University Hospital, New Brunswick, New Jersey
  - Rutgers Cancer Institute of New Jersey-Robert Wood Johnson University Hospital, New Brunswick, New Jersey
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey
  - Rutgers New Jersey Medical School, Newark, New Jersey
  - Newark Beth Israel Medical Center, Newark, New Jersey
  - The Valley Hospital - Luckow Pavilion, Paramus, New Jersey
  - Saint Joseph's Regional Medical Center, Paterson, New Jersey
  - Capital Health Medical Center-Hopewell, Pennington, New Jersey
  - AtlantiCare Regional Medical Center -Main Campus, Pomona, New Jersey
  - Neurosurgeons of New Jersey-Ridgewood, Ridgewood, New Jersey
  - Valley Health System Ridgewood Campus, Ridgewood, New Jersey
  - Sidney Kimmel Cancer Center Washington Township, Sewell, New Jersey
  - Robert Wood Johnson University Hospital Somerset, Somerville, New Jersey
  - Sparta Cancer Treatment Center, Sparta, New Jersey
  - Overlook Hospital, Summit, New Jersey
  - Inspira Medical Center Vineland, Vineland, New Jersey
  - Virtua Voorhees, Voorhees Township, New Jersey
  - Valley Health System-Hematology/Oncology, Westwood, New Jersey
  - Lovelace Medical Center-Saint Joseph Square, Albuquerque, New Mexico
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - Presbyterian Kaseman Hospital, Albuquerque, New Mexico
  - Memorial Medical Center-Las Cruces, Las Cruces, New Mexico
  - Christus Saint Vincent Regional Cancer Center, Santa Fe, New Mexico
  - Maimonides Medical Center, Brooklyn, New York
  - Roswell Park Cancer Institute, Buffalo, New York
  - Memorial Sloan Kettering Commack, Commack, New York
  - Mary Imogene Bassett Hospital, Cooperstown, New York
  - Elmhurst Hospital Center, Elmhurst, New York
  - Arnot Ogden Medical Center/Falck Cancer Center, Elmira, New York
  - Glens Falls Hospital, Glens Falls, New York
  - Memorial Sloan Kettering Westchester, Harrison, New York
  - Queens Hospital Center, Jamaica, New York
  - Northwell Health NCORP, Lake Success, New York
  - Northwell Health/Center for Advanced Medicine, Lake Success, New York
  - North Shore University Hospital, Manhasset, New York
  - Garnet Health Medical Center, Middletown, New York
  - NYU Langone Hospital - Long Island, Mineola, New York
  - Long Island Jewish Medical Center, New Hyde Park, New York
  - Mount Sinai Union Square, New York, New York
  - Laura and Isaac Perlmutter Cancer Center at NYU Langone, New York, New York
  - Mount Sinai West, New York, New York
  - NYP/Columbia University Medical Center/Herbert Irving Comprehensive Cancer Center, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - NYP/Weill Cornell Medical Center, New York, New York
  - Nyack Hospital, Nyack, New York
  - MidHudson Regional Hospital of Westchester Medical Center, Poughkeepsie, New York
  - Rochester General Hospital, Rochester, New York
  - University of Rochester, Rochester, New York
  - Memorial Sloan Kettering Sleepy Hollow, Sleepy Hollow, New York
  - Staten Island University Hospital, Staten Island, New York
  - Stony Brook University Medical Center, Stony Brook, New York
  - State University of New York Upstate Medical University, Syracuse, New York
  - Lincoln Medical and Mental Health Center, The Bronx, New York
  - Montefiore Medical Center-Weiler Hospital, The Bronx, New York
  - Montefiore Medical Center - Moses Campus, The Bronx, New York
  - Memorial Sloan Kettering Nassau, Uniondale, New York
  - Faxton-Saint Luke's Healthcare, Utica, New York
  - Dickstein Cancer Treatment Center, White Plains, New York
  - Atrium Health Stanly/LCI-Albemarle, Albemarle, North Carolina
  - Randolph Hospital, Asheboro, North Carolina
  - Mission Hospital, Asheville, North Carolina
  - Mountain Radiation Oncology PA, Asheville, North Carolina
  - AdventHealth Infusion Center Asheville, Asheville, North Carolina
  - Messino Cancer Centers, Asheville, North Carolina
  - Hope Women's Cancer Centers-Asheville, Asheville, North Carolina
  - Gaston Hematology and Oncology Associates-Belmont, Belmont, North Carolina
  - Transylvania Regional Hospital, Brevard, North Carolina
  - Cone Health Cancer Center at Alamance Regional, Burlington, North Carolina
  - Waverly Hematology Oncology, Cary, North Carolina
  - Carolinas Medical Center/Levine Cancer Institute, Charlotte, North Carolina
  - Novant Health Presbyterian Medical Center, Charlotte, North Carolina
  - Novant Health Carolina Surgical - Randolph, Charlotte, North Carolina
  - Oncology Specialists of Charlotte, Charlotte, North Carolina
  - Atrium Health Pineville/LCI-Pineville, Charlotte, North Carolina
  - Levine Cancer Institute-SouthPark, Charlotte, North Carolina
  - Atrium Health University City/LCI-University, Charlotte, North Carolina
  - Southern Oncology Specialists-Charlotte, Charlotte, North Carolina
  - Levine Cancer Institute-Ballantyne, Charlotte, North Carolina
  - Sampson Radiation Oncology, Clinton, North Carolina
  - Southeastern Medical Oncology Center-Clinton, Clinton, North Carolina
  - Atrium Health Cabarrus/LCI-Concord, Concord, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Cape Fear Valley Health System, Fayetteville, North Carolina
  - Angel Medical Center, Franklin, North Carolina
  - CaroMont Regional Medical Center, Gastonia, North Carolina
  - Gaston Hematology and Oncology Associates, Gastonia, North Carolina
  - Southeastern Medical Oncology Center-Goldsboro, Goldsboro, North Carolina
  - Wayne Memorial Hospital, Goldsboro, North Carolina
  - Wayne Radiation Oncology, Goldsboro, North Carolina
  - Cone Health Cancer Center, Greensboro, North Carolina
  - Maria Parham Hospital, Henderson, North Carolina
  - Margaret R Pardee Memorial Hospital, Hendersonville, North Carolina
  - AdventHealth Hendersonville, Hendersonville, North Carolina
  - Hayworth Cancer Center, High Point, North Carolina
  - High Point Regional Hospital, High Point, North Carolina
  - Novant Health Cancer Institute - Huntersville, Huntersville, North Carolina
  - Southern Oncology Specialists-Huntersville, Huntersville, North Carolina
  - Onslow Memorial Hospital, Jacksonville, North Carolina
  - Southeastern Medical Oncology Center-Jacksonville, Jacksonville, North Carolina
  - ECU Health Oncology Kinston, Kinston, North Carolina
  - Scotland Memorial Hospital-Laurinburg Cancer Center, Laurinburg, North Carolina
  - Novant Health Cancer Institute - Brunswick Forest, Leland, North Carolina
  - Southeastern Regional Medical Center, Lumberton, North Carolina
  - Mission Hospital McDowell, Marion, North Carolina
  - Matthews Radiation Oncology Center, Matthews, North Carolina
  - Novant Health Cancer Institute - Matthews, Matthews, North Carolina
  - Cone Heath Cancer Center at Mebane, Mebane, North Carolina
  - Atrium Health Union/LCI-Union, Monroe, North Carolina
  - Novant Health Cancer Institute - Mooresville, Mooresville, North Carolina
  - Granville Medical Center, Oxford, North Carolina
  - UNC Rex Healthcare, Raleigh, North Carolina
  - Duke Cancer Center Raleigh, Raleigh, North Carolina
  - UNC Rex Cancer Center of Wakefield, Raleigh, North Carolina
  - Annie Penn Memorial Hospital, Reidsville, North Carolina
  - Person Memorial Hospital, Roxboro, North Carolina
  - Rutherford Hospital, Rutherfordton, North Carolina
  - Atrium Health Cleveland/LCI-Cleveland, Shelby, North Carolina
  - Cleveland Hematology and Oncology Associates PC, Shelby, North Carolina
  - Johnston Memorial Hospital, Smithfield, North Carolina
  - Blue Ridge Regional Hospital, Spruce Pine, North Carolina
  - Iredell Memorial Hospital, Statesville, North Carolina
  - Marion L Shepard Cancer Center - ECU Health Beaufort Hospital, Washington, North Carolina
  - Cape Fear Cancer Specialists, Wilmington, North Carolina
  - Novant Health New Hanover Regional Medical Center, Wilmington, North Carolina
  - Southeast Clinical Oncology Research Consortium NCORP, Winston-Salem, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Mid Dakota Clinic, Bismarck, North Dakota
  - Saint Alexius Medical Center, Bismarck, North Dakota
  - Sanford Bismarck Medical Center, Bismarck, North Dakota
  - Altru Cancer Center, Grand Forks, North Dakota
  - Trinity Cancer Care Center, Minot, North Dakota
  - Summa Health System - Akron Campus, Akron, Ohio
  - Cleveland Clinic Akron General, Akron, Ohio
  - Summa Health System - Barberton Campus, Barberton, Ohio
  - Cleveland Clinic Cancer Center Beachwood, Beachwood, Ohio
  - UHHS-Chagrin Highlands Medical Center, Beachwood, Ohio
  - Indu and Raj Soin Medical Center, Beavercreek, Ohio
  - Mary Rutan Hospital, Bellefontaine, Ohio
  - Strecker Cancer Center-Belpre, Belpre, Ohio
  - Toledo Clinic Cancer Centers-Bowling Green, Bowling Green, Ohio
  - Aultman Health Foundation, Canton, Ohio
  - Miami Valley Hospital South, Centerville, Ohio
  - Geauga Hospital, Chardon, Ohio
  - Adena Regional Medical Center, Chillicothe, Ohio
  - Oncology Hematology Care Inc-Eden Park, Cincinnati, Ohio
  - Oncology Hematology Care Inc-Mercy West, Cincinnati, Ohio
  - The Christ Hospital, Cincinnati, Ohio
  - University of Cincinnati Cancer Center-UC Medical Center, Cincinnati, Ohio
  - Good Samaritan Hospital - Cincinnati, Cincinnati, Ohio
  - Oncology Hematology Care Inc-Anderson, Cincinnati, Ohio
  - Oncology Hematology Care Inc-Kenwood, Cincinnati, Ohio
  - Bethesda North Hospital, Cincinnati, Ohio
  - Oncology Hematology Care Inc-Blue Ash, Cincinnati, Ohio
  - TriHealth Cancer Institute-Westside, Cincinnati, Ohio
  - TriHealth Cancer Institute-Anderson, Cincinnati, Ohio
  - Case Western Reserve University, Cleveland, Ohio
  - MetroHealth Medical Center, Cleveland, Ohio
  - Cleveland Clinic Cancer Center/Fairview Hospital, Cleveland, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - North Coast Cancer Care-Clyde, Clyde, Ohio
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - Mount Carmel East Hospital, Columbus, Ohio
  - Columbus Oncology and Hematology Associates Inc, Columbus, Ohio
  - Riverside Methodist Hospital, Columbus, Ohio
  - Columbus NCI Community Oncology Research Program, Columbus, Ohio
  - Grant Medical Center, Columbus, Ohio
  - The Mark H Zangmeister Center, Columbus, Ohio
  - Mount Carmel Health Center West, Columbus, Ohio
  - Doctors Hospital, Columbus, Ohio
  - Grandview Hospital, Dayton, Ohio
  - Good Samaritan Hospital - Dayton, Dayton, Ohio
  - Miami Valley Hospital, Dayton, Ohio
  - Miami Valley Hospital North, Dayton, Ohio
  - Dayton NCI Community Oncology Research Program, Dayton, Ohio
  - Delaware Health Center-Grady Cancer Center, Delaware, Ohio
  - Delaware Radiation Oncology, Delaware, Ohio
  - Grady Memorial Hospital, Delaware, Ohio
  - Hematology Oncology Center Incorporated, Elyria, Ohio
  - Mercy Cancer Center-Elyria, Elyria, Ohio
  - Oncology Hematology Care Inc-Healthplex, Fairfield, Ohio
  - Blanchard Valley Hospital, Findlay, Ohio
  - Atrium Medical Center-Middletown Regional Hospital, Franklin, Ohio
  - Wayne Hospital, Greenville, Ohio
  - Cleveland Clinic Cancer Center Independence, Independence, Ohio
  - First Dayton Cancer Care, Kettering, Ohio
  - Kettering Medical Center, Kettering, Ohio
  - Fairfield Medical Center, Lancaster, Ohio
  - Lancaster Radiation Oncology, Lancaster, Ohio
  - Saint Rita's Medical Center, Lima, Ohio
  - Lima Memorial Hospital, Lima, Ohio
  - OhioHealth Mansfield Hospital, Mansfield, Ohio
  - Cleveland Clinic Cancer Center Mansfield, Mansfield, Ohio
  - Marietta Memorial Hospital, Marietta, Ohio
  - Toledo Clinic Cancer Centers-Maumee, Maumee, Ohio
  - Toledo Radiation Oncology at Northwest Ohio Onocolgy Center, Maumee, Ohio
  - Hillcrest Hospital Cancer Center, Mayfield Heights, Ohio
  - UH Seidman Cancer Center at Landerbrook Health Center, Mayfield Heights, Ohio
  - Summa Health Medina Medical Center, Medina, Ohio
  - UH Seidman Cancer Center at Lake Health Mentor Campus, Mentor, Ohio
  - UH Seidman Cancer Center at Southwest General Hospital, Middleburg Heights, Ohio
  - Knox Community Hospital, Mount Vernon, Ohio
  - Licking Memorial Hospital, Newark, Ohio
  - Newark Radiation Oncology, Newark, Ohio
  - Fisher-Titus Medical Center, Norwalk, Ohio
  - Saint Charles Hospital, Oregon, Ohio
  - Toledo Clinic Cancer Centers-Oregon, Oregon, Ohio
  - University Hospitals Parma Medical Center, Parma, Ohio
  - Mercy Health - Perrysburg Hospital, Perrysburg, Ohio
  - Southern Ohio Medical Center, Portsmouth, Ohio
  - North Coast Cancer Care, Sandusky, Ohio
  - Springfield Regional Cancer Center, Springfield, Ohio
  - Springfield Regional Medical Center, Springfield, Ohio
  - Cleveland Clinic Cancer Center Strongsville, Strongsville, Ohio
  - ProMedica Flower Hospital, Sylvania, Ohio
  - Mercy Hospital of Tiffin, Tiffin, Ohio
  - ProMedica Toledo Hospital/Russell J Ebeid Children's Hospital, Toledo, Ohio
  - Mercy Health - Saint Vincent Hospital, Toledo, Ohio
  - University of Toledo, Toledo, Ohio
  - Toledo Community Hospital Oncology Program CCOP, Toledo, Ohio
  - Mercy Health - Saint Anne Hospital, Toledo, Ohio
  - Toledo Clinic Cancer Centers-Toledo, Toledo, Ohio
  - Upper Valley Medical Center, Troy, Ohio
  - University Hospitals Sharon Health Center, Wadsworth, Ohio
  - South Pointe Hospital, Warrensville Heights, Ohio
  - Fulton County Health Center, Wauseon, Ohio
  - University of Cincinnati Cancer Center-West Chester, West Chester, Ohio
  - Saint Ann's Hospital, Westerville, Ohio
  - UH Seidman Cancer Center at Saint John Medical Center, Westlake, Ohio
  - UHHS-Westlake Medical Center, Westlake, Ohio
  - Clinton Memorial Hospital/Foster J Boyd Regional Cancer Center, Wilmington, Ohio
  - Cleveland Clinic Wooster Family Health and Surgery Center, Wooster, Ohio
  - Wright-Patterson Medical Center, Wright-Patterson Air Force Base, Ohio
  - Greene Memorial Hospital, Xenia, Ohio
  - Genesis Healthcare System Cancer Care Center, Zanesville, Ohio
  - Mercy Clinic Oncology and Hematology-Ardmore, Ardmore, Oklahoma
  - Cancer Centers of Southwest Oklahoma Research, Lawton, Oklahoma
  - Cancer Care Associates-Norman, Norman, Oklahoma
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Mercy Hospital Oklahoma City, Oklahoma City, Oklahoma
  - Mercy Physicians of Oklahoma-Lakeside, Oklahoma City, Oklahoma
  - Natalie Warren Bryant Cancer Center at Saint Francis, Tulsa, Oklahoma
  - Surgical Associates Inc, Tulsa, Oklahoma
  - Oklahoma Cancer Specialists and Research Institute-Tulsa, Tulsa, Oklahoma
  - Warren Clinic Oncology-Tulsa, Tulsa, Oklahoma
  - Saint Alphonsus Cancer Care Center-Baker City, Baker City, Oregon
  - Saint Charles Health System, Bend, Oregon
  - Clackamas Radiation Oncology Center, Clackamas, Oregon
  - Providence Cancer Institute Clackamas Clinic, Clackamas, Oregon
  - Bay Area Hospital, Coos Bay, Oregon
  - Good Samaritan Hospital, Corvallis, Oregon
  - Three Rivers Community Hospital, Grants Pass, Oregon
  - Legacy Mount Hood Medical Center, Gresham, Oregon
  - Asante Health System, Medford, Oregon
  - Asante Rogue Regional Medical Center, Medford, Oregon
  - Providence Medford Medical Center, Medford, Oregon
  - Providence Milwaukie Hospital, Milwaukie, Oregon
  - Providence Newberg Medical Center, Newberg, Oregon
  - Saint Alphonsus Cancer Care Center-Ontario, Ontario, Oregon
  - Providence Willamette Falls Medical Center, Oregon City, Oregon
  - Legacy Good Samaritan Hospital and Medical Center, Portland, Oregon
  - Providence Portland Medical Center, Portland, Oregon
  - Providence Saint Vincent Medical Center, Portland, Oregon
  - Kaiser Permanente Northwest, Portland, Oregon
  - Legacy Emanuel Hospital and Health Center, Portland, Oregon
  - Oregon Health and Science University, Portland, Oregon
  - Legacy Meridian Park Hospital, Tualatin, Oregon
  - Jefferson Abington Hospital, Abington, Pennsylvania
  - Lehigh Valley Hospital-Cedar Crest, Allentown, Pennsylvania
  - UPMC-Heritage Valley Health System Beaver, Beaver, Pennsylvania
  - Saint Luke's University Hospital-Bethlehem Campus, Bethlehem, Pennsylvania
  - Lehigh Valley Hospital - Muhlenberg, Bethlehem, Pennsylvania
  - Bryn Mawr Hospital, Bryn Mawr, Pennsylvania
  - Butler Memorial Hospital, Butler, Pennsylvania
  - Carlisle Regional Cancer Center, Carlisle, Pennsylvania
  - Geisinger Medical Center, Danville, Pennsylvania
  - Doylestown Hospital, Doylestown, Pennsylvania
  - Delaware County Memorial Hospital, Drexel Hill, Pennsylvania
  - Pocono Medical Center, East Stroudsburg, Pennsylvania
  - Easton Hospital, Easton, Pennsylvania
  - Ephrata Cancer Center, Ephrata, Pennsylvania
  - Ephrata Community Hospital, Ephrata, Pennsylvania
  - Adams Cancer Center, Gettysburg, Pennsylvania
  - UPMC Cancer Centers - Arnold Palmer Pavilion, Greensburg, Pennsylvania
  - WellSpan Medical Oncology and Hematology, Hanover, Pennsylvania
  - Geisinger Medical Center-Cancer Center Hazleton, Hazleton, Pennsylvania
  - Penn State Milton S Hershey Medical Center, Hershey, Pennsylvania
  - UPMC-Johnstown/John P. Murtha Regional Cancer Center, Johnstown, Pennsylvania
  - Lancaster General Hospital, Lancaster, Pennsylvania
  - Sechler Family Cancer Center, Lebanon, Pennsylvania
  - Geisinger Medical Oncology-Lewisburg, Lewisburg, Pennsylvania
  - Lewistown Hospital, Lewistown, Pennsylvania
  - UPMC Cancer Center at UPMC McKeesport, McKeesport, Pennsylvania
  - Riddle Memorial Hospital, Media, Pennsylvania
  - UPMC Hillman Cancer Center in Coraopolis, Moon Township, Pennsylvania
  - Suburban Community Hospital and Cancer Center, Norristown, Pennsylvania
  - Paoli Memorial Hospital, Paoli, Pennsylvania
  - Pennsylvania Hospital, Philadelphia, Pennsylvania
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Temple University Hospital, Philadelphia, Pennsylvania
  - Einstein Medical Center Philadelphia, Philadelphia, Pennsylvania
  - Reading Hospital McGlinn Cancer Institute at Phoenixville, Phoenixville, Pennsylvania
  - UPMC-Magee Womens Hospital, Pittsburgh, Pennsylvania
  - UPMC-Presbyterian Hospital, Pittsburgh, Pennsylvania
  - UPMC-Saint Margaret, Pittsburgh, Pennsylvania
  - University of Pittsburgh Cancer Institute (UPCI), Pittsburgh, Pennsylvania
  - UPMC-Shadyside Hospital, Pittsburgh, Pennsylvania
  - UPMC Jefferson Regional Radiation Oncology, Pittsburgh, Pennsylvania
  - UPMC-Passavant Hospital, Pittsburgh, Pennsylvania
  - UPMC-Saint Clair Hospital Cancer Center, Pittsburgh, Pennsylvania
  - Pottstown Hospital, Pottstown, Pennsylvania
  - Geisinger Cancer Services-Pottsville, Pottsville, Pennsylvania
  - Penn State Health Saint Joseph Medical Center, Reading, Pennsylvania
  - Guthrie Medical Group PC-Robert Packer Hospital, Sayre, Pennsylvania
  - Mercy Hospital, Scranton, Pennsylvania
  - Hematology and Oncology Associates of North East Pennsylvania, Scranton, Pennsylvania
  - Scranton Hematology Oncology, Scranton, Pennsylvania
  - Grand View Hospital, Sellersville, Pennsylvania
  - UPMC Cancer Center at UPMC Northwest, Seneca, Pennsylvania
  - Geisinger Medical Group, State College, Pennsylvania
  - Mount Nittany Medical Center, State College, Pennsylvania
  - UPMC Uniontown Hospital Radiation Oncology, Uniontown, Pennsylvania
  - Associates In Hematology Oncology PC-Upland, Upland, Pennsylvania
  - UPMC Washington Hospital Radiation Oncology, Washington, Pennsylvania
  - Chester County Hospital, West Chester, Pennsylvania
  - Reading Hospital, West Reading, Pennsylvania
  - Geisinger Wyoming Valley/Henry Cancer Center, Wilkes-Barre, Pennsylvania
  - UPMC Susquehanna, Williamsport, Pennsylvania
  - Lankenau Medical Center, Wynnewood, Pennsylvania
  - WellSpan Health-York Cancer Center, York, Pennsylvania
  - WellSpan Health-York Hospital, York, Pennsylvania
  - Rhode Island Hospital, Providence, Rhode Island
  - Women and Infants Hospital, Providence, Rhode Island
  - Miriam Hospital, Providence, Rhode Island
  - Roger Williams Medical Center, Providence, Rhode Island
  - Kent Hospital, Warwick, Rhode Island
  - AnMed Health Cancer Center, Anderson, South Carolina
  - AnMed Health Hospital, Anderson, South Carolina
  - Prisma Health Cancer Institute - Spartanburg, Boiling Springs, South Carolina
  - Roper Hospital, Charleston, South Carolina
  - Charleston Oncology - Roper, Charleston, South Carolina
  - Lowcountry Hematology Oncology PA-North Charleston, Charleston, South Carolina
  - Bon Secours Saint Francis Hospital, Charleston, South Carolina
  - Charleston Oncology - Saint Francis, Charleston, South Carolina
  - Lowcountry Hematology Oncology PA-West Ashley, Charleston, South Carolina
  - Medical University of South Carolina, Charleston, South Carolina
  - Prisma Health Cancer Institute - Laurens, Clinton, South Carolina
  - Prisma Health Cancer Institute - Easley, Easley, South Carolina
  - McLeod Regional Medical Center, Florence, South Carolina
  - Gibbs Cancer Center-Gaffney, Gaffney, South Carolina
  - Tidelands Georgetown Memorial Hospital, Georgetown, South Carolina
  - Greenville Health System Cancer Institute-Andrews, Greenville, South Carolina
  - Saint Francis Hospital, Greenville, South Carolina
  - Prisma Health Cancer Institute - Butternut, Greenville, South Carolina
  - Prisma Health Cancer Institute - Faris, Greenville, South Carolina
  - Prisma Health Greenville Memorial Hospital, Greenville, South Carolina
  - Saint Francis Cancer Center, Greenville, South Carolina
  - Prisma Health Cancer Institute - Eastside, Greenville, South Carolina
  - Self Regional Healthcare, Greenwood, South Carolina
  - Prisma Health Cancer Institute - Greer, Greer, South Carolina
  - Gibbs Cancer Center-Pelham, Greer, South Carolina
  - Carolina Blood and Cancer Care Associates PA-Lancaster, Lancaster, South Carolina
  - Lowcountry Hematology Oncology PA-Mount Pleasant, Mt. Pleasant, South Carolina
  - Carolina Blood and Cancer Care Associates PA, Rock Hill, South Carolina
  - Levine Cancer Institute-Rock Hill, Rock Hill, South Carolina
  - Prisma Health Cancer Institute - Seneca, Seneca, South Carolina
  - Spartanburg Medical Center, Spartanburg, South Carolina
  - SMC Center for Hematology Oncology Union, Union, South Carolina
  - Lexington Medical Center, West Columbia, South Carolina
  - Avera Cancer Institute-Aberdeen, Aberdeen, South Dakota
  - Rapid City Regional Hospital, Rapid City, South Dakota
  - Sanford Cancer Center Oncology Clinic, Sioux Falls, South Dakota
  - Avera Cancer Institute, Sioux Falls, South Dakota
  - Medical X-Ray Center, Sioux Falls, South Dakota
  - Avera McKennan Hospital and University Health Center, Sioux Falls, South Dakota
  - Sanford USD Medical Center - Sioux Falls, Sioux Falls, South Dakota
  - Bristol Regional Medical Center, Bristol, Tennessee
  - Wellmont Medical Associates Oncology and Hematology-Bristol, Bristol, Tennessee
  - Erlanger Medical Center, Chattanooga, Tennessee
  - Memorial Hospital, Chattanooga, Tennessee
  - Cookeville Regional Medical Center, Cookeville, Tennessee
  - Vanderbilt-Ingram Cancer Center Cool Springs, Franklin, Tennessee
  - Pulmonary Medicine Center of Chattanooga-Hixson, Hixson, Tennessee
  - Wellmont Medical Associates Oncology and Hematology-Johnson City, Johnson City, Tennessee
  - Ballad Health Cancer Care - Kingsport, Kingsport, Tennessee
  - Wellmont Holston Valley Hospital and Medical Center, Kingsport, Tennessee
  - Thompson Cancer Survival Center, Knoxville, Tennessee
  - University of Tennessee - Knoxville, Knoxville, Tennessee
  - University of Tennessee Health Science Center, Memphis, Tennessee
  - Nashville Breast Center, Nashville, Tennessee
  - Vanderbilt Breast Center at One Hundred Oaks, Nashville, Tennessee
  - Meharry Medical College, Nashville, Tennessee
  - Vanderbilt University/Ingram Cancer Center, Nashville, Tennessee
  - Memorial GYN Plus, Ooltewah, Tennessee
  - The Don and Sybil Harrington Cancer Center, Amarillo, Texas
  - Dell Seton Medical Center at The University of Texas, Austin, Texas
  - Saint Joseph Regional Cancer Center, Bryan, Texas
  - MD Anderson in The Woodlands, Conroe, Texas
  - Dallas VA Medical Center, Dallas, Texas
  - Parkland Memorial Hospital, Dallas, Texas
  - UT Southwestern/Simmons Cancer Center-Dallas, Dallas, Texas
  - Texas Tech University Health Sciences Center-El Paso, El Paso, Texas
  - Baylor All Saints Medical Center at Fort Worth, Fort Worth, Texas
  - University of Texas Medical Branch, Galveston, Texas
  - Lyndon Baines Johnson General Hospital, Houston, Texas
  - Baylor College of Medicine/Dan L Duncan Comprehensive Cancer Center, Houston, Texas
  - Houston Methodist Hospital, Houston, Texas
  - M D Anderson Cancer Center, Houston, Texas
  - MD Anderson West Houston, Houston, Texas
  - Baylor Medical Center at Irving, Irving, Texas
  - Doctor's Hospital of Laredo, Laredo, Texas
  - MD Anderson League City, League City, Texas
  - Covenant Medical Center-Lakeside, Lubbock, Texas
  - UMC Cancer Center / UMC Health System, Lubbock, Texas
  - Texas Tech University Health Sciences Center-Lubbock, Lubbock, Texas
  - Audie L Murphy VA Hospital, San Antonio, Texas
  - Cancer Therapy and Research Center at The UT Health Science Center at San Antonio, San Antonio, Texas
  - University Hospital, San Antonio, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - MD Anderson in Sugar Land, Sugar Land, Texas
  - Scott and White Memorial Hospital, Temple, Texas
  - Blood and Cancer Center of East Texas, Tyler, Texas
  - American Fork Hospital / Huntsman Intermountain Cancer Center, American Fork, Utah
  - Sandra L Maxwell Cancer Center, Cedar City, Utah
  - Logan Regional Hospital, Logan, Utah
  - Intermountain Medical Center, Murray, Utah
  - McKay-Dee Hospital Center, Ogden, Utah
  - Utah Valley Regional Medical Center, Provo, Utah
  - Riverton Hospital, Riverton, Utah
  - Utah Cancer Specialists-Salt Lake City, Salt Lake City, Utah
  - Huntsman Cancer Institute/University of Utah, Salt Lake City, Utah
  - LDS Hospital, Salt Lake City, Utah
  - Saint George Regional Medical Center, St. George, Utah
  - Southwestern Vermont Medical Center, Bennington, Vermont
  - Central Vermont Medical Center/National Life Cancer Treatment, Berlin Corners, Vermont
  - University of Vermont and State Agricultural College, Burlington, Vermont
  - Rutland Regional Medical Center, Rutland, Vermont
  - Ballad Health Cancer Care - Bristol, Bristol, Virginia
  - Kaiser Permanente-Burke Medical Center, Burke, Virginia
  - University of Virginia Cancer Center, Charlottesville, Virginia
  - Sentara Martha Jefferson Hospital, Charlottesville, Virginia
  - Danville Regional Medical Center, Danville, Virginia
  - Fredericksburg Oncology Inc, Fredericksburg, Virginia
  - Hematology Oncology Associates of Fredericksburg Inc, Fredericksburg, Virginia
  - Peninsula Cancer Institute-Gloucester, Gloucester, Virginia
  - Centra Alan B Pearson Regional Cancer Center, Lynchburg, Virginia
  - Kaiser Permanente Tysons Corner Medical Center, McLean, Virginia
  - Peninsula Cancer Institute-Newport News, Newport News, Virginia
  - Ballad Health Cancer Care - Norton, Norton, Virginia
  - VCU Massey Comprehensive Cancer Center, Richmond, Virginia
  - VCU Community Memorial Health Center, South Hill, Virginia
  - Peninsula Cancer Institute-Cancer Specialists of Tidewater, Virginia Beach, Virginia
  - Peninsula Cancer Institute-Williamsburg, Williamsburg, Virginia
  - Providence Regional Cancer System-Aberdeen, Aberdeen, Washington
  - Cancer Care Center at Island Hospital, Anacortes, Washington
  - MultiCare Auburn Medical Center, Auburn, Washington
  - Virginia Mason Bainbridge Island Medical Center, Bainbridge Island, Washington
  - Overlake Medical Center, Bellevue, Washington
  - PeaceHealth Saint Joseph Medical Center, Bellingham, Washington
  - Highline Medical Center-Main Campus, Burien, Washington
  - Providence Regional Cancer System-Centralia, Centralia, Washington
  - Swedish Cancer Institute-Edmonds, Edmonds, Washington
  - Saint Elizabeth Hospital, Enumclaw, Washington
  - Providence Regional Cancer Partnership, Everett, Washington
  - Virginia Mason Federal Way Medical Center, Federal Way, Washington
  - Saint Francis Hospital, Federal Way, Washington
  - Tacoma/Valley Radiation Oncology Centers-Gig Harbor, Gig Harbor, Washington
  - MultiCare Gig Harbor Medical Park, Gig Harbor, Washington
  - Swedish Cancer Institute-Issaquah, Issaquah, Washington
  - Kadlec Clinic Hematology and Oncology, Kennewick, Washington
  - Northwest Cancer Clinic, Kennewick, Washington
  - EvergreenHealth Medical Center, Kirkland, Washington
  - FHCC at EvergreenHealth, Kirkland, Washington
  - Providence Regional Cancer System-Lacey, Lacey, Washington
  - Saint Clare Hospital, Lakewood, Washington
  - PeaceHealth Saint John Medical Center, Longview, Washington
  - Virginia Mason Lynnwood Medical Center, Lynnwood, Washington
  - Skagit Regional Health Cancer Care Center, Mount Vernon, Washington
  - Skagit Valley Hospital, Mount Vernon, Washington
  - Providence - Saint Peter Hospital, Olympia, Washington
  - Capital Medical Center, Olympia, Washington
  - Olympic Medical Center, Port Angeles, Washington
  - Jefferson Healthcare, Port Townsend, Washington
  - Harrison HealthPartners Hematology and Oncology-Poulsbo, Poulsbo, Washington
  - Peninsula Cancer Center, Poulsbo, Washington
  - MultiCare Good Samaritan Hospital, Puyallup, Washington
  - Tacoma/Valley Radiation Oncology Centers-Puyallup, Puyallup, Washington
  - Virginia Mason Medical Center, Seattle, Washington
  - Harborview Medical Center, Seattle, Washington
  - Minor and James Medical PLLC, Seattle, Washington
  - Pacific Gynecology Specialists, Seattle, Washington
  - Pacific Medical Center-First Hill, Seattle, Washington
  - Swedish Medical Center-Ballard Campus, Seattle, Washington
  - Fred Hutchinson Cancer Center, Seattle, Washington
  - Kaiser Permanente Washington, Seattle, Washington
  - Swedish Medical Center-Cherry Hill, Seattle, Washington
  - Swedish Medical Center-First Hill, Seattle, Washington
  - University of Washington Medical Center - Montlake, Seattle, Washington
  - PeaceHealth United General Medical Center, Sedro-Woolley, Washington
  - Olympic Medical Cancer Care Center, Sequim, Washington
  - Providence Regional Cancer System-Shelton, Shelton, Washington
  - Saint Michael Cancer Center, Silverdale, Washington
  - Cancer Care Northwest - Spokane South, Spokane, Washington
  - MultiCare Deaconess Cancer and Blood Specialty Center - Downtown, Spokane, Washington
  - Spokane Valley Cancer Center-Mayfair, Spokane, Washington
  - Cancer Care Northwest-Valley, Spokane, Washington
  - Spokane Valley Cancer Center-Mission, Spokane, Washington
  - Cancer Care Northwest-North Spokane, Spokane, Washington
  - Evergreen Hematology and Oncology PS, Spokane, Washington
  - MultiCare Deaconess Cancer and Blood Specialty Center - North, Spokane, Washington
  - Rockwood Clinic, Spokane, Washington
  - MultiCare Deaconess Cancer and Blood Specialty Center - Valley, Spokane Valley, Washington
  - Tacoma/Valley Radiation Oncology Centers-Jackson Hall, Tacoma, Washington
  - Franciscan Research Center-Northwest Medical Plaza, Tacoma, Washington
  - MultiCare Allenmore Hospital, Tacoma, Washington
  - MultiCare Tacoma General Hospital, Tacoma, Washington
  - Northwest Medical Specialties PLLC, Tacoma, Washington
  - Northwest NCI Community Oncology Research Program, Tacoma, Washington
  - Saint Joseph Medical Center, Tacoma, Washington
  - Tacoma/Valley Radiation Oncology Centers-Saint Joe's, Tacoma, Washington
  - Madigan Army Medical Center, Tacoma, Washington
  - PeaceHealth Southwest Medical Center, Vancouver, Washington
  - Compass Oncology Vancouver, Vancouver, Washington
  - Legacy Salmon Creek Hospital, Vancouver, Washington
  - Providence Saint Mary Regional Cancer Center, Walla Walla, Washington
  - Wenatchee Valley Hospital and Clinics, Wenatchee, Washington
  - North Star Lodge Cancer Center at Yakima Valley Memorial Hospital, Yakima, Washington
  - Providence Regional Cancer System-Yelm, Yelm, Washington
  - United Hospital Center, Bridgeport, West Virginia
  - West Virginia University Charleston Division, Charleston, West Virginia
  - Edwards Comprehensive Cancer Center, Huntington, West Virginia
  - WVUH-Berkely Medical Center, Martinsburg, West Virginia
  - Monongalia Hospital, Morgantown, West Virginia
  - West Virginia University Healthcare, Morgantown, West Virginia
  - Camden Clark Medical Center, Parkersburg, West Virginia
  - Princeton Community Hospital, Princeton, West Virginia
  - Langlade Hospital and Cancer Center, Antigo, Wisconsin
  - ThedaCare Regional Cancer Center, Appleton, Wisconsin
  - ThedaCare Regional Medical Center - Appleton, Appleton, Wisconsin
  - Aurora Cancer Care-Southern Lakes VLCC, Burlington, Wisconsin
  - Marshfield Clinic-Chippewa Center, Chippewa Falls, Wisconsin
  - Marshfield Clinic Cancer Center at Sacred Heart, Eau Claire, Wisconsin
  - Marshfield Medical Center-EC Cancer Center, Eau Claire, Wisconsin
  - Aurora Health Center-Fond du Lac, Fond du Lac, Wisconsin
  - Ascension Saint Francis - Reiman Cancer Center, Franklin, Wisconsin
  - Aurora Health Care Germantown Health Center, Germantown, Wisconsin
  - Aurora Cancer Care-Grafton, Grafton, Wisconsin
  - Green Bay Oncology at Saint Vincent Hospital, Green Bay, Wisconsin
  - Saint Vincent Hospital Cancer Center Green Bay, Green Bay, Wisconsin
  - Saint Vincent Hospital Cancer Center at Saint Mary's, Green Bay, Wisconsin
  - Aurora BayCare Medical Center, Green Bay, Wisconsin
  - Mercyhealth Hospital and Cancer Center - Janesville, Janesville, Wisconsin
  - University of Wisconsin Carbone Cancer Center - Johnson Creek, Johnson Creek, Wisconsin
  - Aurora Cancer Care-Kenosha South, Kenosha, Wisconsin
  - Gundersen Lutheran Medical Center, La Crosse, Wisconsin
  - Mayo Clinic Health System-Franciscan Healthcare, La Crosse, Wisconsin
  - University of Wisconsin Carbone Cancer Center - University Hospital, Madison, Wisconsin
  - Holy Family Memorial Hospital, Manitowoc, Wisconsin
  - Aurora Bay Area Medical Group-Marinette, Marinette, Wisconsin
  - Bay Area Medical Center, Marinette, Wisconsin
  - Marshfield Medical Center-Marshfield, Marshfield, Wisconsin
  - Ascension Columbia Saint Mary's Hospital Ozaukee, Mequon, Wisconsin
  - Aurora Cancer Care-Milwaukee, Milwaukee, Wisconsin
  - Ascension Southeast Wisconsin Hospital - Saint Joseph Campus, Milwaukee, Wisconsin
  - Ascension Columbia Saint Mary's Hospital - Milwaukee, Milwaukee, Wisconsin
  - Aurora Saint Luke's Medical Center, Milwaukee, Wisconsin
  - Medical College of Wisconsin, Milwaukee, Wisconsin
  - Aurora Sinai Medical Center, Milwaukee, Wisconsin
  - Marshfield Medical Center - Minocqua, Minocqua, Wisconsin
  - ProHealth D N Greenwald Center, Mukwonago, Wisconsin
  - Cancer Center of Western Wisconsin, New Richmond, Wisconsin
  - ProHealth Oconomowoc Memorial Hospital, Oconomowoc, Wisconsin
  - Saint Vincent Hospital Cancer Center at Oconto Falls, Oconto Falls, Wisconsin
  - Vince Lombardi Cancer Clinic - Oshkosh, Oshkosh, Wisconsin
  - Ascension All Saints Hospital, Racine, Wisconsin
  - Aurora Cancer Care-Racine, Racine, Wisconsin
  - Aspirus Cancer Care - James Beck Cancer Center, Rhinelander, Wisconsin
  - Marshfield Medical Center-Rice Lake, Rice Lake, Wisconsin
  - HSHS Saint Nicholas Hospital, Sheboygan, Wisconsin
  - Vince Lombardi Cancer Clinic-Sheboygan, Sheboygan, Wisconsin
  - Aspirus Cancer Care - Stevens Point, Stevens Point, Wisconsin
  - Marshfield Medical Center-River Region at Stevens Point, Stevens Point, Wisconsin
  - Saint Vincent Hospital Cancer Center at Sturgeon Bay, Sturgeon Bay, Wisconsin
  - Aurora Medical Center in Summit, Summit, Wisconsin
  - Vince Lombardi Cancer Clinic-Two Rivers, Two Rivers, Wisconsin
  - Aurora Cancer Care-Waukesha, Waukesha, Wisconsin
  - ProHealth Waukesha Memorial Hospital, Waukesha, Wisconsin
  - UW Cancer Center at ProHealth Care, Waukesha, Wisconsin
  - Aspirus Regional Cancer Center, Wausau, Wisconsin
  - Marshfield Clinic-Wausau Center, Wausau, Wisconsin
  - Aurora Cancer Care-Milwaukee West, Wauwatosa, Wisconsin
  - Aurora West Allis Medical Center, West Allis, Wisconsin
  - Marshfield Medical Center - Weston, Weston, Wisconsin
  - Aspirus Cancer Care - Wisconsin Rapids, Wisconsin Rapids, Wisconsin
  - Marshfield Clinic - Wisconsin Rapids Center, Wisconsin Rapids, Wisconsin
  - Rocky Mountain Oncology, Casper, Wyoming
  - Cheyenne Regional Medical Center-West, Cheyenne, Wyoming
  - Big Horn Basin Cancer Center, Cody, Wyoming
  - Billings Clinic-Cody, Cody, Wyoming
  - Welch Cancer Center, Sheridan, Wyoming
- Canada (28):
  - BCCA-Abbotsford Cancer Centre, Abbotsford, British Columbia
  - BCCA-Cancer Centre for the Southern Interior, Kelowna, British Columbia
  - BCCA-Fraser Valley Cancer Centre, Surrey, British Columbia
  - BCCA-Vancouver Cancer Centre, Vancouver, British Columbia
  - CancerCare Manitoba, Winnipeg, Manitoba
  - Atlantic Health Sciences Corporation-Saint John Regional Hospital, Saint John, New Brunswick
  - Doctor H. Bliss Murphy Cancer Centre, St. John's, Newfoundland and Labrador
  - Royal Victoria Regional Health Centre, Barrie, Ontario
  - Health Sciences North, Greater Sudbury, Ontario
  - Juravinski Cancer Centre at Hamilton Health Sciences, Hamilton, Ontario
  - Waterloo Regional Health Network, Kitchener, Ontario
  - Trillium Health Partners - Credit Valley Hospital, Mississauga, Ontario
  - Thunder Bay Regional Health Science Centre, Thunder Bay, Ontario
  - Michael Garron Hospital, Toronto, Ontario
  - Mount Sinai Hospital, Toronto, Ontario
  - University Health Network-Princess Margaret Hospital, Toronto, Ontario
  - Trillium Health Partners - Queensway Health Centre, Toronto, Ontario
  - PEI Cancer Treatment Centre-Queen Elizabeth Hospital, Charlottetown, Prince Edward Island
  - CIUSSSEMTL-Hopital Maisonneuve-Rosemont, Montreal, Quebec
  - McGill University Department of Oncology, Montreal, Quebec
  - CHUM-Hotel Dieu de Montreal, Montreal, Quebec
  - CHUM - Centre Hospitalier de l'Universite de Montreal, Montreal, Quebec
  - The Research Institute of the McGill University Health Centre (MUHC), Montreal, Quebec
  - Jewish General Hospital, Montreal, Quebec
  - CHU de Quebec-Hopital du Saint-Sacrement (HSS), Québec, Quebec
  - Centre Hospitalier Universitaire de Sherbrooke-Fleurimont, Sherbrooke, Quebec
  - Allan Blair Cancer Centre, Regina, Saskatchewan
  - Saskatoon Cancer Centre, Saskatoon, Saskatchewan
- Instituto Nacional De Cancerologia, Bogotá, Colombia
- France (59):
  - Institut de Cancerologie de l'Ouest- Angers, Angers
  - Centre Hospitalier d'Auch, Auch
  - Institut Sainte Catherine, Avignon
  - Centre d'Oncologie et de Radiotherapie Pays Basque, Bayonne
  - Centre Hospitalier de la Cote Basque, Bayonne
  - Centre Hospitalier de Beauvais, Beauvais
  - Centre Hospitalier de Blois, Blois
  - Clinique Tivoli Ducos, Bordeaux
  - Institut Bergonie Cancer Center, Bordeaux
  - Polyclinic Bordeaux Nord Aquitaine, Bordeaux
  - CHU de Brest-Hopital Morvan, Brest
  - Centre Francois Baclesse, Caen
  - Centre Jean Perrin, Clermont-Ferrand
  - Centre Hospitlier Intercommunal de Creteil, Créteil
  - Centre Hospitalier de Douai, Dechy
  - Centre Georges-Francois Leclerc, Dijon
  - Hopital Prive Drome Ardeche-Clinique Pasteur, Guilherand-Granges
  - Departemental Hospitalier Roche-sur-Yon (Les Oudairies), La Roche-sur-Yon
  - Hopital Prive de l'Estuaire, Le Havre
  - Clinique Victor Hugo-Centre Jean Bernard, Le Mans
  - Centre Oscar Lambert, Lille
  - Clinique Chenieux, Limoges
  - CHU Limoges - Hopital Dupuytren, Limoges
  - Hopital Prive Jean Mermoz, Lyon
  - Centre Leon Berard, Lyon
  - Hopital Prive Clairval, Marseile
  - Centre Hospitalier de Montelimar, Montélimar
  - Centre Catherine de Sienne, Nantes
  - Clinique Hartmann, Neuilly-sur-Seine
  - Centre Antoine Lacassagne, Nice
  - Hospital De La Source, Orléans
  - Institut Curie Paris, Paris
  - Hopital Saint Louis, Paris
  - Hopital Prive des Peupliers, Paris
  - Hôpital La Pitié-Salpétrière, Paris
  - Centre Hopitalier, Pau
  - Clinical Saint-Pierre/Centre Catalan d?Oncologie, Perpignan
  - Centre Hospitalier de Perpignan, Perpignan
  - Polyclinique Francheville, Périgueux
  - Centre hospitalier Rene Dubos Pontoise, Pontoise
  - Institut Jean Godinot, Reims
  - Centre Henri Becquerel, Rouen
  - Institut Curie-Centre Rene Huguenin Saint Cloud, Saint-Cloud
  - Centre Hospitalier Prive Saint-Gregoire, Saint-Grégoire
  - Institut de Cancerologie de l'Ouest-Rene Gauducheau, Saint-Herblain
  - Clinique Mutualiste de l'Estuaire, Saint-Nazaire
  - Centre de Cancerologie Paris Nord, Sarcelles
  - Groupe Hospitalier Public du Sud de l'Oise Senlis, Senlis
  - Centre Paul Strauss, Strasbourg
  - CHRU Strasbourg - Hospital Civil, Strasbourg
  - Polyclinique de l'Ormeau, Tarbes
  - Hopitaux du Leman, Thonon-les-Bains
  - Center Claudius Regaud, Toulouse
  - Clinique Pasteur, Toulouse
  - Clinique Saint-Jean Languedoc, Toulouse
  - Hospital Bretonneau, Tours
  - Centre Alexis Vautrin, Vandœuvre-lès-Nancy
  - Gustave Roussy, Villejuif
  - Hopital Prive de Villeneuve d'Ascq, Villeneuve
- Ireland (14):
  - Bon Secours Hospital, Cork, Co Cork
  - Tallaght University Hospital, Dublin, Co Dublin
  - Saint Vincent's University Hospital, Dublin, Co Dublin
  - Mater Misericordiae University Hospital, Dublin, Co Dublin
  - Mater Private Hospital, Dublin, Co Dublin
  - Beaumont Hospital, Dublin, Co Dublin
  - Saint Vincent's Private Hospital, Mount Merrion, Co Dublin
  - University College Hospital Galway, Galway, Co Galway
  - Mid-Western Regional Hospital, Limerick, Co Limerick
  - Sligo University Hospital, Sligo, Co Sligo
  - University Hospital Waterford, Waterford, Co Waterford
  - Cork University Hospital, Cork
  - Saint James Hospital, Dublin
  - Letterkenny General Hospital, Letterkenny
- Instituto Nacional De Cancerologia de Mexico, Mexico City, Tlalpan, Mexico
- Puerto Rico (4):
  - Cancer Center-Metro Medical Center Bayamon, Bayamón
  - Doctors Cancer Center, Manatí
  - San Juan Community Oncology Group, San Juan
  - San Juan City Hospital, San Juan
- King Faisal Specialist Hospital and Research Centre, Riyadh, Saudi Arabia
- South Korea (3):
  - National Cancer Center-Korea, Goyang-si, Gyeonggi-do
  - Seoul National University Bundang Hospital, Seongnam, Kyeonggi-do
  - Asan Medical Center, Seoul
- Spain (22):
  - Centro Oncologico de Galicia, A Coruña
  - Complejo Hospitalario Universitario de Albacete, Albacete
  - Hospital De La Santa Creu I Sant Pau, Barcelona
  - Hospital Clinic De Barcelona, Barcelona
  - Hospital Universitari Germans Trias i Pujol, Barcelona
  - Hospital Provincial de Castellon, Castellon
  - Hospital San Pedro de Alcantara, Cáceres
  - Hospital Nuestra Senora de Aranzazu, Donostia / San Sebastian
  - Onkologikoa, Donostia / San Sebastian
  - Grupo Espanol de Investigacion en Cancer de Mama, Donostia / San Sebastian
  - Institut Catalad'Oncologia, Girona
  - Hospital Universitari de Girona Doctor Josep Trueta, Girona
  - Hospital Universitario Gregorio Maranon, Madrid
  - Hospital Universitario Ramon y Cajal, Madrid
  - Hospital Infanta Cristina de Parla, Madrid
  - Hospital Clinico Universitario Virgen de la Victoria, Málaga
  - Hospital Universitario Virgen del Rocio, Seville
  - Hospital Virgen de la Salud, Toledo
  - Instituto Valenciano de Oncologia, Valencia
  - Hospital Clinico Universitario de Valencia, Valencia
  - Hospital Clinico Universitario Lozano Blesa, Zaragoza
  - Hospital Universitario Miguel Servet, Zaragoza

REFERENCES:
- [Derived] Kang IM, Forschmiedt JK, Loch MM, Lew DL, Barlow WE, Gralow JR, Meric-Bernstam F, Albain KS, Hayes DF, Lin NU, Perez EA, Goldstein LJ, Rastogi P, Schott AF, Baehner R, Sharma P, Tripathy D, Pusztai L, Hortobagyi GN, Kalinsky K, Henry NL. Cognitive Impairment and Chemoendocrine vs Endocrine Therapy in Pre- and Postmenopausal Women: A Secondary Analysis of the RxPONDER Randomized Clinical Trial. JAMA Oncol. 2025 Dec 11:e255220. doi: 10.1001/jamaoncol.2025.5220. Online ahead of print. PMID 41379459
- [Derived] Abdou Y, Barlow WE, Gralow JR, Meric-Bernstam F, Albain KS, Hayes DF, Lin NU, Perez EA, Goldstein LJ, Chia SKL, Dhesy-Thind S, Rastogi P, Alba E, Delaloge S, Schott AF, Shak S, Sharma P, Lew DL, Miao J, Unger JM, Tripathy D, Hortobagyi GN, Pusztai L, Kalinsky K. Race and clinical outcomes in hormone receptor-positive, HER2-negative, node-positive breast cancer in the randomized RxPONDER trial. J Natl Cancer Inst. 2025 May 1;117(5):889-897. doi: 10.1093/jnci/djae314. PMID 39656951
- [Derived] Kalinsky K, Barlow WE, Gralow JR, Meric-Bernstam F, Albain KS, Hayes DF, Lin NU, Perez EA, Goldstein LJ, Chia SKL, Dhesy-Thind S, Rastogi P, Alba E, Delaloge S, Martin M, Kelly CM, Ruiz-Borrego M, Gil-Gil M, Arce-Salinas CH, Brain EGC, Lee ES, Pierga JY, Bermejo B, Ramos-Vazquez M, Jung KH, Ferrero JM, Schott AF, Shak S, Sharma P, Lew DL, Miao J, Tripathy D, Pusztai L, Hortobagyi GN. 21-Gene Assay to Inform Chemotherapy Benefit in Node-Positive Breast Cancer. N Engl J Med. 2021 Dec 16;385(25):2336-2347. doi: 10.1056/NEJMoa2108873. Epub 2021 Dec 1. PMID 34914339

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 9383 participants were screened and 5083 were randomized to the trial: 2547 to the Chemo and Endocrine Therapy arm and 2536 to the Endocrine Therapy Alone arm. In the Chemo and Endocrine Therapy Arm, 36 were ineligible. In the Endocrine Therapy Alone arm, 29 were ineligible. Ultimately, 5018 participants were eligible in the participant flow: 2511 in the Chemo and Endocrine Therapy arm and 2507 in the Endocrine Therapy Alone arm.
Groups:
- Chemo and Endocrine Therapy: Participants receive a protocol-approved chemotherapy regimen based on the participant and/or physician preference. Participants then receive a protocol-approved adjuvant endocrine therapy for 5-10 years in the absence of disease progression or unacceptable toxicity.
- Endocrine Therapy Alone: Participants receive a protocol-approved endocrine therapy for 5-10 years in the absence of disease progression or unacceptable toxicity.
Period: Overall Study
Arm/Group | Chemo and Endocrine Therapy | Endocrine Therapy Alone
Started | 2511 | 2507
Completed | 1504 | 1547
Not Completed | 1007 | 960
Not completed — Death | 25 | 28
Not completed — Adverse Event | 12 | 7
Not completed — Withdrawal by Subject | 175 | 93
Not completed — Disease progression | 70 | 111
Not completed — Other reason | 42 | 41
Not completed — Delinquent data | 24 | 19
Not completed — Reason under review | 33 | 29
Not completed — On treatment | 626 | 632

BASELINE CHARACTERISTICS:
Population: Randomized participants who were eligible for the study.
Groups:
- Total: Total of all reporting groups
Arm/Group | Chemo and Endocrine Therapy | Endocrine Therapy Alone | Total
Number analyzed (Participants) | 2511 | 2507 | 5018
Age, Continuous [Median (Full Range); unit: years] | 57.9 [28.0 to 87.6] | 57.2 [18.3 to 86.0] | 57.5 [18.3 to 87.6]
Age, Customized [Count of Participants; unit: Participants]
  < 40 years | 67 | 80 | 147
  40-49 years | 530 | 547 | 1077
  50-59 years | 837 | 838 | 1675
  60-69 years | 777 | 761 | 1538
  >= 70 years | 300 | 281 | 581
Sex: Female, Male [Count of Participants; unit: Participants] — This trial only included female participants.
  Participants
    Female | 2511 | 2507 | 5018
    Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 297 | 325 | 622
  Not Hispanic or Latino | 1731 | 1695 | 3426
  Unknown or Not Reported | 483 | 487 | 970
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 1667 | 1628 | 3295
  Black | 130 | 121 | 251
  Asian | 154 | 170 | 324
  Other/Unknown | 560 | 588 | 1148
Menopausal Status [Count of Participants; unit: Participants] — Premenopausal was defined as: < 6 months since last menstrual period and no prior bilateral oophorectomy and not on estrogen replacement.
  Postmenopausal was defined as: prior bilateral oophorectomy, or > 12 months since last menstrual period with no prior hysterectomy.
  If these categories did not apply, premenopausal was defined as age < 50 and postmenopausal was defined as age >= 50.
  Participants
    Premenopausal | 834 | 831 | 1665
    Postmenopausal | 1677 | 1676 | 3353
Recurrence Score [Count of Participants; unit: Participants] — The Oncotype DX® Recurrence Score is based on a 21-gene breast cancer assay. The score ranges from 0-100, with higher scores indicating a worse prognosis. This study included participants with a score of 0-25.
  Participants
    0-13 | 1076 | 1071 | 2147
    14-25 | 1435 | 1436 | 2871
Axillary Surgery [Count of Participants; unit: Participants]
  Axillary lymph-node dissection, with or without sentinel-node mapping | 1569 | 1571 | 3140
  Sentinel-node biopsy without axillary lymph-node dissection | 942 | 936 | 1878
Positive Nodes [Count of Participants; unit: Participants]
  1 node | 1628 | 1647 | 3275
  2 nodes | 643 | 623 | 1266
  3 nodes | 231 | 229 | 460
  Not reported | 9 | 8 | 17

OUTCOME MEASURES:

1. Primary Outcome: Invasive Disease-Free Survival (IDFS)
Description: From date of randomization (2nd Registration) to date of first invasive recurrence (local, regional or distant), second invasive primary cancer (breast or not), or death due to any cause. Patients last known to be alive who have not experienced recurrence or second primary cancer are censored at their last contact date. This is the STEEP definition of invasive disease-free survival. Kaplan-Meier estimates were calculated for the 5-year IDFS rate.
  Due to the results of the third prespecified interim analysis, prespecified separate analyses were conducted for all outcomes by menopausal status (see Statistical Analysis 2). The NCI and data and safety monitoring committee recommended early reporting of the data. After the primary analysis, changes in eligibility status were identified for three participants, making the population of eligible and evaluable participants different between the reporting of this outcome and both the Participant Flow section and the Adverse Events section.
Time Frame: 5 years after randomization
Population: For the participants flow and baseline characteristics summary, 5018 eligible participants were included. However, among them, there were 34 participants (10 in the chemo and endocrine arm, and 24 in the endocrine alone arm) that withdrew consent immediately after randomization; thus these participants were excluded from the survival analyses.
Measure: Number; unit: percentage of participants
Arm/Group | Chemo and Endocrine Therapy | Endocrine Therapy Alone
Number analyzed (Participants) | 2487 | 2497
percentage of participants
  Premenopausal: number analyzed (Participants) | 829 | 826
  Premenopausal | 93.9 | 89.0
  Postmenopausal: number analyzed (Participants) | 1658 | 1671
  Postmenopausal | 91.3 | 91.9
Statistical Analysis 1: Comparison: Chemo and Endocrine Therapy vs Endocrine Therapy Alone; This test describes the interaction of the treatment arm with the recurrence score in the analysis of invasive disease-free survival in the overall study population, to determine whether chemotherapy benefit depends on the recurrence score. If the interaction was statistically significant, the interaction term was planned to be included in the Cox model to evaluate the invasive disease-free survival outcome; Test type: Other; p = 0.35, Regression, Cox; A Cox model was used that included treatment arm, recurrence score, menopausal status, and the chemotherapy*recurrence score interaction term; Hazard Ratio (HR) = 1.02, 95% CI 2-sided [0.98 to 1.05]
Statistical Analysis 2: Comparison: Chemo and Endocrine Therapy vs Endocrine Therapy Alone; This test describes the interaction of the treatment arm with menopausal status (one of the study stratification factors) in the analysis of invasive disease-free survival in the overall study population, to determine whether chemotherapy benefit depends on menopausal status. If the interaction was statistically significant, separate analyses of IDFS were planned to be conducted by menopausal status; Test type: Other; p = 0.008, Regression, Cox; A Cox model was used that included treatment arm, recurrence score, menopausal status, and the chemotherapy*menopausal status interaction term; Hazard Ratio (HR) = 1.71, 95% CI 2-sided [1.15 to 2.54]
Statistical Analysis 3: Comparison: Chemo and Endocrine Therapy vs Endocrine Therapy Alone; This analysis includes only premenopausal participants; Test type: Superiority; p = 0.002, Regression, Cox; Hazard Ratio (HR) = 0.60, 95% CI 2-sided [0.43 to 0.83] — To compare the Chemo and Endocrine Therapy arm to the Endocrine Therapy Alone arm, a Cox model was used with adjustment for the continuous recurrence score
Statistical Analysis 4: Comparison: Chemo and Endocrine Therapy vs Endocrine Therapy Alone; This analysis includes only postmenopausal participants; Test type: Superiority; p = 0.89, Regression, Cox; Hazard Ratio (HR) = 1.02, 95% CI 2-sided [0.82 to 1.26] — [estimate comment as in outcome 1, analysis 3]

2. Secondary Outcome: Number of Participants With Gr 3 Through 5 Adverse Events That Are Related to Study Drugs
Description: Only adverse events that are possibly, probably, or definitely related to study drug are reported. Assessed at 6, 12, 24, and 36 months after randomization.
Time Frame: Duration of treatment and follow-up until death or 3 years after randomization
Population: Eligible participants who received at least one dose of protocol treatment and assessed for Adverse Event.
Measure: Number; unit: Participants
Arm/Group | Chemo and Endocrine Therapy | Endocrine Therapy Alone
Number analyzed (Participants) | 2062 | 2342
Participants
  Abdominal infection | 1 | 0
  Abdominal pain | 7 | 0
  Acute kidney injury | 1 | 0
  Alanine aminotransferase increased | 4 | 2
  Alkaline phosphatase increased | 1 | 0
  Allergic reaction | 6 | 1
  Anemia | 20 | 0
  Anorexia | 2 | 0
  Anxiety | 2 | 1
  Arthralgia | 48 | 35
  Aspartate aminotransferase increased | 0 | 1
  Atrial fibrillation | 3 | 1
  Back pain | 1 | 1
  Blood and lymphatic system disorders - Other | 4 | 0
  Bone marrow hypocellular | 1 | 0
  Bone pain | 15 | 5
  Breast infection | 2 | 0
  Bronchial infection | 1 | 0
  CD4 lymphocytes decreased | 2 | 1
  Cardiac arrest | 1 | 0
  Cataract | 0 | 1
  Catheter related infection | 3 | 0
  Chest pain - cardiac | 1 | 0
  Chest wall pain | 0 | 1
  Colitis | 5 | 0
  Constipation | 4 | 0
  Death NOS | 0 | 1
  Dehydration | 11 | 0
  Depression | 3 | 6
  Dermatitis radiation | 4 | 4
  Device related infection | 4 | 0
  Diarrhea | 31 | 3
  Dizziness | 3 | 1
  Dry mouth | 1 | 0
  Dry skin | 1 | 0
  Dyspareunia | 1 | 1
  Dyspepsia | 1 | 0
  Dyspnea | 2 | 0
  Ear pain | 2 | 0
  Edema limbs | 1 | 0
  Ejection fraction decreased | 1 | 0
  Erythema multiforme | 1 | 0
  Erythroderma | 1 | 1
  Esophagitis | 3 | 0
  Fatigue | 48 | 9
  Febrile neutropenia | 83 | 1
  Fever | 3 | 0
  Flank pain | 1 | 0
  Flu like symptoms | 1 | 0
  GGT increased | 2 | 0
  Gastric hemorrhage | 1 | 0
  Gastric ulcer | 1 | 0
  Gastrointestinal disorders - Other, specify | 1 | 0
  Gastrointestinal pain | 1 | 0
  General disorders and admin site conditions - Other | 2 | 0
  Generalized muscle weakness | 4 | 0
  Headache | 7 | 1
  Heart failure | 1 | 0
  Hematuria | 1 | 0
  Hemorrhoids | 1 | 0
  Hot flashes | 12 | 14
  Hyperglycemia | 16 | 1
  Hyperhidrosis | 1 | 0
  Hypertension | 8 | 6
  Hypokalemia | 5 | 0
  Hyponatremia | 2 | 0
  Hypotension | 3 | 1
  INR increased | 0 | 1
  Infections and infestations - Other, specify | 3 | 0
  Injection site reaction | 1 | 0
  Insomnia | 9 | 4
  Irregular menstruation | 3 | 1
  Joint range of motion decreased | 1 | 0
  Kidney infection | 1 | 0
  Left ventricular systolic dysfunction | 1 | 0
  Leukemia secondary to oncology chemotherapy | 2 | 0
  Leukocytosis | 4 | 0
  Lipase increased | 1 | 0
  Localized edema | 1 | 1
  Lung infection | 6 | 0
  Lymphedema | 1 | 1
  Lymphocyte count decreased | 20 | 0
  Menorrhagia | 0 | 1
  Mucositis oral | 23 | 0
  Muscle weakness lower limb | 1 | 0
  Musculoskeletal and connective tiss disorder - Other | 1 | 0
  Myalgia | 24 | 8
  Myelitis | 1 | 0
  Myocardial infarction | 2 | 0
  Nausea | 21 | 0
  Neck pain | 2 | 0
  Neoplasms benign, malignant and unspecified - Other | 3 | 0
  Nervous system disorders - Other, specify | 1 | 0
  Neutrophil count decreased | 150 | 1
  Osteoporosis | 1 | 0
  Pain | 2 | 0
  Pain in extremity | 2 | 1
  Palmar-plantar erythrodysesthesia syndrome | 7 | 0
  Paresthesia | 2 | 0
  Peripheral ischemia | 0 | 1
  Peripheral motor neuropathy | 4 | 0
  Peripheral sensory neuropathy | 21 | 2
  Platelet count decreased | 3 | 0
  Pleuritic pain | 1 | 0
  Pneumonitis | 8 | 0
  Premature menopause | 1 | 0
  Pruritus | 5 | 1
  Radiation recall reaction (dermatologic) | 2 | 0
  Rash acneiform | 1 | 0
  Rash maculo-papular | 8 | 2
  Renal and urinary disorders - Other, specify | 1 | 0
  Reproductive system and breast disorders - Other | 1 | 0
  Sepsis | 5 | 0
  Sinus tachycardia | 1 | 0
  Skin and subcutaneous tissue disorders - Other | 6 | 5
  Skin infection | 9 | 0
  Skin ulceration | 1 | 0
  Stroke | 2 | 3
  Suicidal ideation | 1 | 0
  Supraventricular tachycardia | 1 | 1
  Surgical and medical procedures - Other, specify | 2 | 4
  Syncope | 3 | 0
  Thromboembolic event | 9 | 4
  Tinnitus | 1 | 0
  Typhlitis | 1 | 0
  Upper gastrointestinal hemorrhage | 1 | 0
  Upper respiratory infection | 1 | 0
  Urinary tract infection | 4 | 0
  Urticaria | 4 | 0
  Uterine hemorrhage | 0 | 1
  Vaginal dryness | 0 | 4
  Vaginal hemorrhage | 1 | 1
  Vascular access complication | 1 | 0
  Vomiting | 19 | 0
  Watering eyes | 4 | 0
  Weight gain | 4 | 1
  Weight loss | 2 | 0
  White blood cell decreased | 65 | 0
  Wound dehiscence | 1 | 0

3. Secondary Outcome: Overall Survival (OS)
Description: Time from date of randomization (2nd Registration) to date of death due to any cause. Participants last known to be alive are censored at their last contact date.
Time Frame: 5.5 years after randomization
Reporting Status: Not Posted, anticipated posting 2026-12

4. Secondary Outcome: Distant Disease-Free Survival (DDFS)
Description: Time from date of randomization (2nd Registration) to date of invasive distant disease recurrence, second invasive primary cancer (breast or not) or death due to any cause. Participants last known to be alive who have not experienced distant recurrence, or second primary cancer are censored at their last contact date. This secondary outcome requires continuing to follow the patient after local recurrence in order to ascertain subsequent distant recurrence.
  Invasive recurrence is defined as: appearance of any new invasive lesion(s) during or after protocol treatment. Whenever possible, recurrences should be documented histologically. Invasive recurrence includes local, regional, or distant recurrence with an invasive component. A new diagnosis of ipsilateral or contralateral DCIS without an invasive component is not considered to be a recurrence.
Time Frame: 5.5 years after randomization
Reporting Status: Not Posted, anticipated posting 2026-12

5. Secondary Outcome: Local Disease-Free Interval (LDFI)
Description: Time from date of randomization (2nd Registration) to date of invasive local or regional recurrence. Participants last known to be alive without recurrence are censored at their last contact date. Participants with distant recurrence, second primary cancer or death are censored at the time of that event.
  Invasive recurrence is defined as: appearance of any new invasive lesion(s) during or after protocol treatment. Whenever possible, recurrences should be documented histologically. Invasive recurrence includes local, regional, or distant recurrence with an invasive component. A new diagnosis of ipsilateral or contralateral DCIS without an invasive component is not considered to be a recurrence.
Time Frame: From date of randomization to a maximum of 5.5 years or death
Reporting Status: Not Posted, anticipated posting 2026-12

6. Secondary Outcome: Participant-Reported Anxiety
Description: Anxiety is evaluated with the Patient-Reported Outcomes Measurement Information System (PROMIS) Emotional Distress-Anxiety Short Form. Raw PROMIS scores can be re-scaled into T-scores based on a reference population with a mean score of 50 and a standard deviation of 10. Higher scores reflect greater anxiety.
  PROMIS Anxiety scores at the 6 month timepoint will be compared between the two randomized study arms separately by menopausal status.
Time Frame: 6 months after randomization
Reporting Status: Not Posted, anticipated posting 2026-12

7. Secondary Outcome: Participant-Reported Health Status
Description: Assessed using the EuroQol-5D (EQ-5D), in which participants rate their health status in five different health-related domains: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. The raw scores can be converted to index scores on a scale of 0 to 1, where a higher index score represents better health.
  EQ-5D index scores at the 6-month timepoint will be compared between the two randomized study arms separately by menopausal status.
Time Frame: 6 months after randomization
Reporting Status: Not Posted, anticipated posting 2026-12

8. Post Hoc Outcome: Distant Relapse-Free Survival (DRFS)
Description: Time from date of randomization (2nd Registration) to date of invasive distant disease recurrence or death due to any cause. Participants last known to be alive who have not experienced distant recurrence are censored at their last contact date. This outcome requires continuing to follow the patient after local recurrence in order to ascertain subsequent distant recurrence. Kaplan-Meier estimates were calculated for the 5-year DRFS rate.
  Due to the results of the third prespecified interim analysis, prespecified separate analyses were conducted for all outcomes by menopausal status. The NCI and the data and safety monitoring committee recommended early reporting of the data. Due to subsequent data collection and data cleaning, the population of eligible and evaluable participants differs slightly between the reporting of this outcome and the Participant Flow section.
Time Frame: 5 years after randomization
Population: Eligible and evaluable participants
Measure: Number; unit: percentage of participants
Arm/Group | Chemo and Endocrine Therapy | Endocrine Therapy Alone
Number analyzed (Participants) | 2487 | 2497
percentage of participants
  Premenopausal participants: number analyzed (Participants) | 829 | 826
  Premenopausal participants | 96.1 | 92.8
  Postmenopausal participants: number analyzed (Participants) | 1658 | 1671
  Postmenopausal participants | 94.4 | 94.4
Statistical Analysis 1: Comparison: Chemo and Endocrine Therapy vs Endocrine Therapy Alone; This analysis includes only premenopausal participants; Test type: Superiority; p = 0.009, Regression, Cox; Hazard Ratio (HR) = 0.58, 95% CI 2-sided [0.39 to 0.87]; To compare DRFS between the Chemo and Endocrine Therapy arm and the Endocrine Therapy Alone arm, a Cox model was used with adjustment for the continuous recurrence score
Statistical Analysis 2: Comparison: Chemo and Endocrine Therapy vs Endocrine Therapy Alone; This analysis includes only postmenopausal participants; Test type: Superiority; p = 0.70, Regression, Cox; Hazard Ratio (HR) = 1.05, 95% CI 2-sided [0.81 to 1.37] — To compare DRFS between the Chemo and Endocrine Therapy arm and the Endocrine Therapy Alone arm, a Cox model was used with adjustment for the continuous recurrence score

ADVERSE EVENTS:
Time Frame: Adverse Events were assessed for the duration of treatment and follow-up until death or 3 years after randomization. All-Cause Mortality was assessed up to 5 years from randomization. CTCAE Version 4.0 was used for routine toxicity reporting. Version 5.0 was used for Serious Adverse Event (SAE) reporting.
Description: Only participants who received protocol treatment and assessed for adverse event were included in the adverse event result: 2062 in the Chemo and Endocrine Therapy arm and 2342 in the Endocrine Therapy Alone arm.
  All-Cause mortality is reported for all eligible and evaluable participants (2487 in the Chemo and Endocrine arm and 2497 in the endocrine therapy arm). Due to eligibility changes found after the primary analysis, the number at risk differs from the Outcomes Section.
Arm/Group | Chemo and Endocrine Therapy | Endocrine Therapy Alone
All-Cause Mortality (participants affected / at risk) | 161/2487 | 175/2497
Serious Adverse Events (participants affected / at risk) | 14/2062 | 9/2342
Other Adverse Events (participants affected / at risk) | 151/2062 | 2/2342
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Chemo and Endocrine Therapy (N=2062) | Endocrine Therapy Alone (N=2342)
Anemia (Blood and lymphatic system disorders) | 1 | 0
Cardiac arrest (Cardiac disorders) | 2 | 2
Gastrointestinal disorders-Other (Gastrointestinal disorders) | 1 | 0
Typhlitis (Gastrointestinal disorders) | 1 | 0
Upper gastrointestinal hemorrhage (Gastrointestinal disorders) | 1 | 0
Death NOS (General disorders) | 1 | 1
Multi-organ failure (General disorders) | 0 | 1
Device related infection (Infections and infestations) | 1 | 0
Sepsis (Infections and infestations) | 3 | 0
Injury, poison and procedural complications - Other (Injury, poisoning and procedural complications) | 1 | 0
Leukemia secondary to oncology chemotherapy (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Neoplasms benign, malignant and unspecified - Other (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Stroke (Nervous system disorders) | 0 | 3
Pregnancy, puerperium and perinatal conditions-Other (Pregnancy, puerperium and perinatal conditions) | 0 | 1
Thromboembolic event (Vascular disorders) | 2 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Chemo and Endocrine Therapy (N=2062) | Endocrine Therapy Alone (N=2342)
Neutrophil count decreased (Investigations) | 151 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-12-10): https://cdn.clinicaltrials.gov/large-docs/37/NCT01272037/Prot_SAP_000.pdf